

# PM1183-A-018-20

An Open-Label, Multicenter Study to Assess the Potential Effects of Itraconazole (a Strong CYP3A4 Inhibitor) on the Pharmacokinetics of Lurbinectedin (PM01183) in Patients with Advanced Solid Tumors

STATISTICAL ANALYSIS PLAN

INVESTIGATIONAL MEDICINAL PRODUCTS: Lurbinectedin and Itraconazole

Protocol Code: PM1183-A-018-20 EudraCT No: 2020-001332-96 NCT Code: NCT05063318

Version: v2.0

Date: 27-MAY-2022

# TABLE OF CONTENTS

| 1 | | ' RATIONALE | _ |
|---|---|---|---|
| 2 | OVER/ | ALL STUDY DESIGN | 6 |
| 3 | PATIE | NTS EVALUABILITY CRITERIA | 9 |
| 4 | STUDY | OBJECTIVES AND PHARMACOKINETIC PARAMETERS | . 10 |
| | | ectives | |
| | 4.1.1 | Primary | |
| | 4.1.2 | Secondary | |
| | 4.1 End | lpoints | |
| | 4.1.1 | Primary | |
| | 4.1.2 | Secondary | |
| 5 | | LE CONSIDERATIONS | |
| • | | adomization | |
| | | nple Size | |
| 6 | | STICAL METHODOLOGY | |
| Ü | | ricity and Adverse Events | |
| | | nical Laboratory Evaluation | |
| | | rsical Examination, Vital signs, Left Ventricular Ejection Fraction and | . 12 |
| | | diogram Findings | 13 |
| | | oths and other Serious Adverse Events | |
| 7 | | ANALYSES | |
| , | | lent Disposition and Treatment/Study Discontinuation | |
| | | tocol Deviations | |
| | | eline and Demographic Data | |
| | | atment Administration | |
| | | sequent Therapies | |
| | | outation in Incomplete Dates | |
| | | iable Unit Standardization | |
| | | cimal Places, Missing Values and Allowed Assessment Windows | |
| | | egroup Analyses | |
| | 7.9 Suc<br>7.10 | Pharmacogenetic Analysis | |
| | 7.10 | Identification of Fixed or Random Effects Models | |
| | 7.11 | Data Analysis Conventions | |
| 8 | | • | |
| - | | | |
| | | or superior will be used for all statistical analysis outputs | |
| 9 | | ENCES DIX I: PATIENTS DISPOSITION | |
| 1( | | | |
| | 10.1 | General Characteristics | |
| | 10.1.1 | Patient Disposition | |
| | 10.1.2 | Treatment Discontinuations | |
| | 10.1.3 | Protocol Deviations | |
| | 10.2 | Patient Characteristics | |
| | 10.2.1 | Demographic and Other Baseline Characteristics | |
| | 10.2.2 | Medical History | |
| | 10.2.3 | Cancer History | |
| | 10.2.4 | Previous Anticancer Therapy Summary | |
| | 10.2.5 | Physical Examination, ECOG, Vital Signs, LVEF and ECG | |
| | 10.2.6 | Hematological Evaluation at Baseline | . 30 |

| 10.2.7 | Biochemical Evaluation at Baseline | 31 |
|----------|------------------------------------------------------|----|
| 10.2.8 | Coagulation Evaluation at Baseline | 32 |
| 10.2.9 | Signs and Symptoms at Baseline | 33 |
| 10.2.10 | Concomitant Medication at Baseline | 35 |
| 11 APPEN | DIX II: SAFETY ANALYSIS | 36 |
| 11.1 | Extent of Exposure | 36 |
| 11.1.1 | Treatment Administration | 36 |
| 11.1.2 | Cycle Delays | 37 |
| 11.1.3 | Dose Reductions | |
| 11.1.4 | Any Other Dose Modifications | 39 |
| 11.2 | Adverse Events (AEs) | |
| 11.2.1 | Display of Adverse Events | 40 |
| 11.2.2 | Evolution of Signs and Symptoms during the Treatment | 49 |
| 11.3 | Serious Adverse Events and Deaths | 50 |
| 11.3.1 | Serious Adverse Events | 50 |
| 11.3.2 | Deaths | 54 |
| 11.4 | Clinical Laboratory Evaluation | 55 |
| 11.4.1 | Hematological Abnormalities | 55 |
| 11.4.2 | Biochemical Abnormalities | 57 |
| 11.4.3 | Laboratory Values Over Treatment | 59 |
| 11.5 | Linear Mixed-effects Model | 61 |
| 11.6 | Physical Findings, ECOG PS, LVEF and ECG | 62 |
| 11.6.1 | Physical Findings and ECOG PS | 62 |
| 11.6.2 | LVEF and ECG | 62 |
| 11.7 | Concomitant Therapies | 65 |
| 11.7.1 | Concomitant Medication during the Study | 65 |
| | Further Antitumor Therapies | |
| 12 APPEN | DIX III: EFFICACY EVALUATION | 67 |
| 13 APPEN | DIX IV: DB Listings | 68 |
| 14 APPEN | DIX V: BIMO Listings | 73 |
| | DIX VI: ICH Listings | |
| 15.1 | History of Changes | 76 |

#### ABBREVIATIONS AND GLOSSARY

**AE(s)** Adverse Event(s)

ALT Alanine Aminotransferase
AST Aspartate Aminotransferase

ATC Anatomical Therapeutic Chemical

**AUC** Area Under the Concentration-time Curve

BIMO Bioresearch Monitoring
BSA Body Surface Area
CI Confidence Interval

**Cl** Clearance

C<sub>max</sub> Maximum Plasma Concentration

**CPK** Creatine Phosphokinase

**CPK-MB** Creatine Phosphokinase Isoenzyme MB

CrCl Creatinine Clearance
CRF Case Report Form
CRP C-reactive Protein
CV Coefficient of Variation
CYP Cytochrome P450

**D** Day

**DL** Dose Level

DSBs Double-strand Breaks
ECG Electrocardiogram
ECHO Echocardiogram

**ECOG PS** Eastern Cooperative Oncology Group Performance Status

**EDC** Electronic Data Capture

**EOT** End of treatment

**FDA** Food and Drug Administration

GCP Good Clinical Practice
GGT Gamma-glutamyltransferase

HR Heart Rate

IC Informed Consent

IC50 Half Maximal Inhibitory ConcentrationICH International Conference on Harmonization

IEC Independent Ethics CommitteeINR International Normalized RatioIRB Institutional Review Board

i.v. Intravenous

L Liter

**LDH** Lactate Dehydrogenase

LRB Lurbinectedin

**LVEF** Left Ventricular Ejection Fraction

**MedDRA** Medical Dictionary for Regulatory Activities

MinMinutesMgMilligrammLMilliliter

MUGA Multiple-gated Acquisition Scan

NA Not Applicable

**NCI-CTCAE** National Cancer Institute Common Toxicity Criteria

**PD** Progressive Disease

PGt Pharmacogenetic
PK Pharmacokinetics
PN Preferred Name
PS Performance Status
PT Preferred Term
q3wk Every Three Weeks
Pandomized

R Randomized RBC Red Blood Cells

**RT** Reference-Test Sequence

**RTSM** Randomization and Trial Supply Management

S Sequence

SAE(s)Serious Adverse Event(s)SAPStatistical Analysis PlanSCLCSmall Cell Lung Cancer

**SmPC** Summary of Product Characteristics

SOC System Organ Class T<sub>1/2</sub> Terminal Half-life

**TEAE(s)** Treatment-Emergent Adverse Events

TR Test-Reference Sequence ULN Upper Limit of Normal

Vs. Versus

Vss Volume of Distribution at Steady State

**WBC** White Blood Cells

WHO World Health Organization

wk Week(s)

#### 1 STUDY RATIONALE

Lurbinectedin (PM01183) is a novel synthetic tetrahydroisoquinoline structurally related to ecteinascidins.

Lurbinectedin is a new chemical entity that binds the DNA leading to the formation of DNA double-strand breaks (DSBs). The binding to DNA is likely occurring in the minor groove region and induces apoptosis and delayed progression through the cellular phase S/G2. Lurbinectedin also induces the specific degradation of transcribing RNA Pol II in several human tumor cell lines.

In vitro, lurbinectedin demonstrated cytotoxic effects against a broad selection of tumor types with half maximal inhibitory concentration (IC50) values in the range of 1-10 nM. Although selectivity was also seen, a clustering of sensitive tumors has not been identified. Lurbinectedin also exhibited antitumor activity against different murine models of xenografted human-derived tumor types. Lurbinectedin has been tested as a single agent or in combination with different drugs in solid tumors; while antitumor activity in hematological tumors was deemed negligible, lurbinectedin has shown activity in different solid tumors; some of the most responsive tumor types were breast, small cell lung cancer (SCLC), ovarian and endometrial cancer.

Based on current clinical data, the toxicity of lurbinectedin is predictable, reversible and manageable. The most relevant toxicity is reversible myelosuppression with a nadir occurring in the middle of the second week after Day 1 infusion in an every-three-week cycle; overall, the incidence of febrile neutropenia is below 20% in all ongoing Phase II trials.

Lurbinectedin is extensively metabolized by the cytochrome P450 enzymes, primarily CYP3A4. Thus, potent inducers or inhibitors of this enzyme may alter the plasma concentrations of lurbinectedin. This study is designed to examine the pharmacokinetics (PK) and safety of lurbinectedin when co-administered with itraconazole, a strong CYP3A4 inhibitor, in comparison with lurbinectedin alone. The results of this study may be used to support future clinical studies in patients and prescribing information in future labeling.

A full rationale for the study may be found in the appropriate sections of the study's clinical protocol.

#### 2 OVERALL STUDY DESIGN

This is a prospective, open-label, two-way crossover, phase Ib drug-drug interaction study in patients with advanced solid tumors.

The study will include a pre-treatment (screening) phase (within 14 days before the first lurbinectedin or itraconazole administration) followed by a treatment phase consisting of two lurbinectedin cycles, one cycle in combination with itraconazole and one cycle of lurbinectedin as single agent (in different order depending on the study sequence), and one additional third cycle of lurbinectedin as a single agent for patients who meet the continuation criteria and obtain a clinical benefit after the first two cycles, and then follow-up of adverse events if any.

Patients who meet the continuation criteria and obtain a clinical benefit according to the Investigator's criteria will have the opportunity to continue treatment under a Compassionate Use Agreement after the completion of the optional third study cycle.

Patients will be treated as outpatients. At the discretion of the Investigator, patients may be admitted to the study center on Day -1 or Day 1 and monitored, at least, until completion of the Day 1 PK blood sample collections.

Patients will receive a maximum of three cycles: two consecutive cycles of lurbinectedin, one cycle with and one cycle without itraconazole co-administration (in different order depending on the study Sequence 1 or Sequence 2 of treatment), followed by a third cycle with lurbinectedin alone (this last optional for patients with clinical benefit). Lurbinectedin will be administered as a 1-hour (-5/+20 min) i.v. infusion q3wk via a central or peripheral vein.

In the co-administration cycles, itraconazole will be administered orally once daily in the morning after breakfast during 12 consecutive days, self-administered at home from Day -4 (i.e., four days before lurbinectedin infusion) until Day 8 (i.e., seven days after lurbinectedin infusion), and supplied at the study center on Day 1, following recommendations at the Summary of Product Characteristics (SmPC). On Day 1 (i.e., the day of lurbinectedin infusion), itraconazole will be given immediately prior to starting the lurbinectedin infusion. In fact, itraconazole should be administered after obtain the itraconazole PK sample #1 and before the start of lurbinectedin infusion (-15 min to -1 min).

In case of lurbinectedin delay ( $\leq 2$  days), itraconazole could be administered during a maximum of 14 days.

This study will consist of two parts: Part A and B. The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A will be 0.8 mg/m², and in Part B is susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A. The dose of lurbinectedin during Parts A and B will be 3.2 mg/m² for all patients when administered without itraconazole. If toxicity occurs, the appropriate intra-patient dose level (DL) reductions will be implemented in the subsequent cycle.



In Part A, three patients will be enrolled to Sequence 1 (TR: Test-Reference) and will receive itraconazole with lurbinectedin in Cycle 1 followed by two consecutive cycles of lurbinectedin alone (the last cycle being optional for patients with clinical benefit according to the Investigator's criteria).

Enrollment for Part A will be sequential. Once the first patient enrolled has completed Cycle 1 and Cycle 2, the second and the third patients could be enrolled simultaneously, after the evaluation of lurbinected ntotal PK parameters, and if no unacceptable or lifethreatening toxicities have occurred for this first patient. However, if toxicity occurs, the

appropriate dose reductions will be implemented with the second and third patients based on the PK and safety information of first patient.

The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A will be 0.8 mg/m<sup>2</sup>. However, if lurbinectedin exposure in the first patient of Part A does not allow an adequate PK assessment, the lurbinectedin dose of the following patients may be increased accordingly.

Upon exposure and safety assessments in Part A, the dose of lurbinectedin to be co-administered with itraconazole in Part B can be readjusted accordingly. This decision will be made by the Sponsor and study Investigators, and will be documented and communicated to the Independent Ethics Committee/Institutional Review Board (IEC/IRB).

Therefore, the planned dose of lurbinectedin, when given with itraconazole for the remaining eight patients in Part B will be based on the acceptability of the PK and safety results from the first three patients in Part A. If the initial three patients do not experience adverse events (AEs) which might require a dose reduction, the dose of lurbinectedin may still be adjusted (based on the assumption of dose-proportional PK) to produce plasma lurbinectedin AUC values that are comparable to those when lurbinectedin is given in the absence of itraconazole. However, if toxicity occurs in the initial three patients in Part A, the appropriate dose-reduction of lurbinectedin will be implemented in Part B accordingly.

If the safety and PK data obtained from the three patients in Part A is deemed acceptable as defined in the protocol, Part B of this study will begin enrollment. Therefore, once Part A is completed, patients in Part B will be enrolled based on the review of the safety following completion of the first cycle of the previous patient(s), and will be randomized in a 1:1 ratio to Sequence 1 (as used in Part A) or Sequence 2 (RT: Reference-Test; lurbinectedin + itraconazole in Cycle 2).

In Part A, all patients will receive itraconazole plus lurbinectedin in Cycle 1 and lurbinectedin alone in Cycles 2 and 3 (this last cycle being optional).

In Part B, patients will be randomly assigned to the corresponding sequences:

- Sequence 1 (TR) (same used in Part A):
  - o Cycle 1: Itraconazole + lurbinectedin
  - o Cycle 2: Lurbinectedin alone
  - o Cycle 3: Lurbinectedin alone (optional)
- Sequence 2 (RT):
  - o Cycle 1: Lurbinectedin alone
  - o Cycle 2: Itraconazole + lurbinectedin
  - o Cycle 3: Lurbinectedin alone (optional)

Lurbinectedin will be administered to 11 evaluable patients for PK analyses and for a maximum of three cycles, while considered to be on the patient's best interest or until PD, unacceptable toxicity, intercurrent illness of sufficient magnitude to preclude safe continuation of the study, patient's refusal and/or non-compliance with study requirements, a protocol deviation with an effect on the risk/benefit ratio of the clinical

study, more than one lurbinectedin dose reduction due to AEs related to lurbinectedin (unless clear clinical benefit has been documented and always with the Sponsor's agreement) or any other reason at the physician's judgment that precludes lurbinectedin continuation.

If the patient responds to treatment after the first two cycles, treatment with lurbinectedin may continue outside this study under a Compassionate Use Agreement at the same dose based on Investigator's decision and upon agreement with the Sponsor. Then, the treating center must request authorization to the relevant Health Authorities and notify the Sponsor in due time. In order to avoid a treatment discontinuation, during the Compassionate Use Agreement authorization an additional third cycle with lurbinectedin is allowed.

All adverse events (AEs) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5. Treatment delays, dose reduction requirements and reasons for treatment discontinuation will be monitored throughout the study. The safety profile of patients will be monitored throughout the treatment and up to 31 days (±10 days) after the last lurbinectedin infusion (end of treatment, EOT), until the patient starts a new antitumor therapy or until the date of death, whichever occurs first. Any treatment-emergent AEs will be followed until recovery to at least grade 1 or stabilization of symptoms or until the start of a new antitumor therapy, until the continuation of treatment outside this study under a Compassionate Use Agreement or death, whichever occurs first. After treatment discontinuation, patients will be followed until resolution or stabilization of all toxicities, if any.

Patients will be evaluated at scheduled visits on three study periods: pre-treatment (screening), treatment (one cycle of lurbinectedin in combination with itraconazole and two as a single agent and the third cycle optional) and follow-up of adverse events if any.

#### 3 PATIENTS EVALUABILITY CRITERIA

Patients must fulfill all the inclusion/exclusion criteria to be eligible to participate in the study.

The study will include the following analysis population set definitions:

- The <u>enrolled population</u> is defined as all patients recorded in the database who are included in the trial, independently of whether they have received the study drug or not. Screening failure patients will not be considered as part of this population.
- The <u>PK population</u> will include all patients enrolled in Part A and B who have sufficient and interpretable PK parameters to calculate the non-compartmental PK parameters. Only the patients in Part B who have completed the two cycles and have sufficient and interpretable PK assessments will be included in the statistical comparison to assess the effect of itraconazole on the PK of lurbinectedin.
- The <u>safety population</u> will include all patients who received at least one dose of lurbinectedin. Patients who have received at least one dose of itraconazole but who did not receive any dose of lurbinectedin will be excluded from the safety population. The analysis of data from these patients will be performed separately (e.g., by means of narratives). The safety population will be used for all safety evaluations.

# 4 STUDY OBJECTIVES AND PHARMACOKINETIC PARAMETERS

#### 4.1 Objectives

This clinical pharmacology study is designed to assess the impact of itraconazole coadministration on lurbinectedin PK parameters administered alone.

#### 4.1.1 Primary

• To assess the effect of itraconazole on lurbinectedin total plasma exposure in patients with advanced solid tumors.

#### 4.1.2 Secondary

- To assess the effect of itraconazole on lurbinectedin unbound plasma exposure.
- To assess the effect of itraconazole on lurbinectedin major metabolites (i.e., M1 and M4).
- To assess the effect of itraconazole on the safety profile of lurbinectedin.
- To collect and store a blood sample for germline DNA extraction for future pharmacogenetic (PGt) analysis of variations on genes that may influence exposure and response (i.e., disposition, metabolism and safety) to lurbinectedin.

#### 4.1 Endpoints

#### 4.1.1 Primary

• Plasma dose-normalized  $C_{max}$  and  $AUC_{0-\infty}$  of lurbinectedin will be compared between Cycle 1 and Cycle 2. Pharmacokinetic analyses will be evaluated in plasma by standard non-compartmental methods, or population methods, if necessary.

#### 4.1.2 Secondary

- Differences in dose-normalized total AUC<sub>0-t</sub> and Cmax and in Cl, Vss and T<sub>1/2</sub> of lurbinectedin between Cycle 1 and Cycle 2 will be explored.
- Differences in dose-normalized unbound  $AUC_{u,0}-\infty$ ,  $AUC_{u,0-t}$  and  $C_{u,max}$  and in  $CL_u$ , Vss,u and  $T_{1/2},u$  of lurbinectedin between Cycle 1 and Cycle 2 will be explored.
- Differences in ratios between total AUC<sub>0-∞</sub>, AUC0-t and Cmax, of main lurbinectedin metabolites relative to parent drug between Cycle 1 and Cycle 2 will be explored. Additional PK parameters will be calculated if deemed appropriate.
- Treatment safety, including AEs, serious adverse events (SAEs) and laboratory abnormalities will be graded according to the NCI-CTCAE v.5. Additionally, treatment compliance, in particular dose reductions requirements and/or treatment delays due to AEs, and reasons for treatment discontinuation will also be described. Patients will be evaluable for safety if they have received at least one partial or complete infusion of lurbinectedin.

• The presence or absence of PGt polymorphisms in genes relevant for lurbinectedin disposition (distribution, metabolism and excretion) from a single blood sample collected (only if written IC given) at any time during the trial (but preferably at the same time as the pre-treatments PK sample on Day 1 of Cycle 1), which will be stored to explain individual variability in main PK parameters in future analyses

#### 5 SAMPLE CONSIDERATIONS

#### 5.1 Randomization

A block randomization (1:1 ratio) will be performed only in Part B. Block randomization will be used to avoid bias in the assignment of patients to treatment sequence group, to increase the likelihood that known and unknown subject attributes (e.g., demographic and baseline characteristics) are evenly balanced across treatment sequence groups, and to enhance the validity of statistical comparisons across treatment sequence groups.

Patients must be replaced if they are not evaluable for the assessment of the primary endpoint (e.g., if they have not sufficient and interpretable PK parameters).

An evaluable patient for Part A should have completed sufficient study procedures until Day 8 of Cycle 1 (i.e., most itraconazole administration and PK assessments). For Part B, an evaluable patient for the main objective of the study (e.g., assessment of lurbinectedin PK) should have provided sufficient and interpretable PK parameters (e.g.,  $AUC_{0-t}$  should cover at least 80% of  $AUC_{0-\infty}$ ) of Cycle 1 and 2. Evaluable patients should have received the first two complete cycles regardless dose delays or reductions. For Part A and Part B, the compliance of itraconazole will be confirmed based on a patient's diary, the drug accountability and the expected individual plasma concentration at the steady state.

Randomization will be implemented in Medidata Rave RTSM for Part B of the study. A randomization list will be generated to randomly allocate patients to the sequence treatment. Additional randomization lists will be generated in case non-evaluable patients need to be replaced. Variable block sizes and allocation ratios will be used depending on the number of patients to be replaced in each case scenario in order to complete both sequence treatment groups while keeping balance across them. In order to achieve reproducible results, the seed used in the generation of each randomization list will be saved.

#### 5.2 Sample Size

This study was designed to assess the potential effects of itraconazole on the PK of lurbinectedin in patients with advanced malignancies. The 90% CI will be used to help with the interpretation of the results. A sample size of eight patients was based on feasibility and clinical considerations. Based on previous studies, the intra-subject coefficient of variation (CV) of lurbinectedin PK parameters is estimated to be more than 30%. The precision (half-width) of the 90% CI for [(lurbinectedin + itraconazole) / lurbinectedin alone] comparison on the log-scale will extend 0.389 from the observed differences in means, assuming that the intra-subject CV around 40%. This half-width corresponds to a 90% CI in the range of 70% and 147% assuming the ratio of the means equal to unity for each PK parameter. This 90% CI will be used to help with the interpretation of the results.

#### 6 STATISTICAL METHODOLOGY

The PK definitions and analysis plan will be described by the Pharmacology department in a separate document. The present SAP is focused on the statistical methodology for safety.

Safety analyses will consider treatment emergent AEs and SAEs, according to their relationship with study treatment, as well as analytical results, deaths and the reasons for treatment discontinuations, delays and/or dose reductions. All AEs and SAEs will be graded according to NCI-CTCAE v.5, and coded using the Medical Dictionary for Regulatory Activities (MedDRA).

Descriptive statistics will be used to characterize the profiles of drug-related AEs, drug-related deaths, SAEs, clinical laboratory data, drug-related delays and/or treatment discontinuations. Tables will be displayed by study part and sequence of treatment (Test/Reference or Reference/Test).

## 6.1 Toxicity and Adverse Events

Treatment-emergent adverse events (TEAEs) are any adverse event aggravated in severity from baseline or having their onset between the first dose of the study drug and 31-day ( $\pm 10$  days) after the last treatment dose, death or date of further therapy, whichever came first. AEs related to the study treatment or with unknown relationship occurring more than 31 days after the last dose were also taken into account as TEAEs.

Summary of overall AEs will be done by system organ class (SOC) and preferred term (PT), by severity (worst toxicity grade) and by relationship to the study drug (any of them or both). Tables will be sorted by category of events using SOC (i.e. alphabetic order) and PT in descending frequencies (i.e. from higher to lower).

AEs, SAEs, deaths, laboratory evaluations, dose delays/omissions/reductions and study drug discontinuations due to AEs will be tabulated in a descriptive way. Counts and percentages will be used for categorical variables, and summary tables will be used for continuous variables.

Patients having any treatment-related grade  $\geq 3$  AEs should have relevant tests reassessed at least every 72 hours until recovery to at least grade 2.

#### 6.2 Clinical Laboratory Evaluation

Laboratory results will be classified according to the NCI-CTCAE v.5. All laboratory visits reported as "End of treatment" visit will be mapped to the last cycle visit for each patient.

The following hematological values will be displayed: white blood cells count (WBC), neutrophil count, lymphocyte count, monocyte count, erythrocytes, hemoglobin, hematocrit and platelet count. Worst grade per patient and per cycle for anaemia, lymphopenia, neutropenia, leukopenia and thrombocytopenia during treatment will be shown.

Overall cross tabulation will be presented for the worst grade during treatment vs. the baseline toxicity grading of anaemia, lymphopenia, neutropenia, leukopenia and thrombocytopenia.

If a grade 3/4 neutropenia or thrombocytopenia increase occurs during a treatment cycle, the first day the onset value is reached (counting from the start of the cycle) will be tabulated. Time to recovery of the abnormality (i.e., grade 3/4 neutropenia or thrombocytopenia) will be assessed and defined as the time, in days, from the start of the grade 3/4 abnormality until the abnormality is recovered (grade  $\leq 2$ ). The analysis will be carried out taking into account all events, including those that occur in a same cycle. The information will be shown by means of median and range.

Likewise, the following biochemical and coagulation values will be displayed: aspartate aminotransferase (AST), alanine aminotransferase (ALT), lactate dehydrogenase (LDH), creatinine, creatinine clearance, glucose, creatine phosphokinase (CPK), CPK-MB fraction, gamma glutamyltransferase (GGT), total bilirubin, direct bilirubin, serum electrolytes (Na+, K+, Mg++, Ca++), total proteins, albumin, C-reactive protein count (CRP) and the international normalized ratio (INR). Worst grade per patient and per cycle for applicable values during treatment will be shown.

Time to recovery of the abnormality (grade 3/4 AST or ALT) will be assessed and defined as the time, in days, from the start of the grade 3/4 abnormality until recovery to grade  $\leq$  2. The analysis will be carried out taking into account all events, including those that occur in a same cycle. The information will be shown by means of median and range.

Overall cross tabulation will be presented for the worst grade during treatment vs. the baseline toxicity grading of biochemical abnormalities.

# 6.3 Physical Examination, Vital signs, Left Ventricular Ejection Fraction and Electrocardiogram Findings

Summary tables will be prepared with the performance status, physical examination, body weight and BSA, vital signs, left ventricular ejection fraction (LVEF) and electrocardiogram (ECG) abnormalities. If appropriate, a "change from baseline" summary will also be done.

ECG will be collected in triplicate allowing rhythm definition (at least 30 seconds of duration), PR interval and QT interval (raw and corrected by HR using Bazett's formula). Mean of all ECGs collected on each time point will be used for analysis.

#### 6.4 Deaths and other Serious Adverse Events

Serious adverse events (SAEs) will be tabulated following the same pattern than AEs. Reason of death will be tabulated. In addition, all deaths within 60 days from the first dose of treatment or within 30 days from the last dose of treatment will be listed.

#### 7 OTHER ANALYSES

Continuous variables will be tabulated and presented with summary statistics (i.e., mean, StD, median and range).

Categorical variables will be summarized in frequency tables by means of counts and percentages. Percentages in the summary tables will be rounded and may therefore not always add up to exactly 100%.

## 7.1 Patient Disposition and Treatment/Study Discontinuation

The number of patients included in the study, the number of patients treated and the number of patients evaluable for the main endpoint will be shown. Also, accrual by center and the main dates of the study will be displayed. Reasons for treatment discontinuation and for study discontinuation will be tabulated.

#### 7.2 Protocol Deviations

Protocol deviations will be listed and categorized according to the following categories:

- Inclusion/exclusion criteria not met
- Incorrect treatment, dose or schedule received
- Excluded concomitant medication received
- Withdrawal criteria met, but treatment continued
- Failure to comply study procedures
- Any other Ethical/GCP issues

In addition, they will be classified as Relevant/Non-relevant according to clinical criteria.

## 7.3 Baseline and Demographic Data

Baseline data such as demographics, cancer history, prior therapy, prior relevant history, signs and symptoms, electrocardiogram, LVEF, physical examination, vital signs, laboratory values and concomitant medication, coded according to the World Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) classification system, will be described following standard tables detailed in Appendix I.

Age, baseline weight, height and BSA values will be summarized descriptively. Age categories, sex, race and baseline ECOG PS score will be summarized with frequency counts.

For the cancer history, time from initial diagnosis, time from metastatic disease, time from locally advanced disease and time from last progression before the study entry will be summarized. This time calculations will be shown in months and summarized descriptively. Tumor type and other characteristics of the primary and current disease will be described using standard tables detailed in Appendix I.

Previous relevant medical history (other than cancer) will be listed.

A frequency tabulation of the number of patients with the different types of previous surgery, radiotherapy or therapy (number of lines) will be given.

Signs and symptoms will be displayed by tabulation of frequencies according to NCI-CTCAE v.5 toxicity grades. Signs and symptoms will be listed.

In case of pre-treatment characteristics with multiple measurements per subject before the start of treatment (e.g. laboratory assessments or vital signs), the last value prior to or on the first day of treatment will be considered the baseline measurement.

#### 7.4 Treatment Administration

Exposure to treatment will be described by sequence treatment group.

Total cumulative dose, time on treatment, dose intensity and relative dose intensity, administration delay and dose reductions/omissions will be described following standard

tables (detailed in Section 11, Appendix II). The reported cycle information on the case report form (CRF) pages will be used for the analysis.

Time on treatment, expressed in weeks, is defined as the last administration date of lurbinectedin minus the first administration date of lurbinectedin plus 31 days, except if the patient dies or starts a new antitumor therapy within 31 days from the last administration date, in which case the time on treatment will be the date of death or the start date of the new antitumor therapy minus the date of the first administration of the study treatment.

Total cumulative dose by drug, expressed in mg for both lurbinectedin and itraconazole, is the sum of all the product doses received during the study, including the dose received in the last cycle.

For lurbinectedin, intended dose intensity is the planned dose per cycle divided by the planned number of weeks by cycle.

Absolute dose intensity is the actual cumulative dose divided by the number of weeks of treatment. As a convention, for this calculation, the duration of the last cycle will be the predefined cycle length (e.g, 21 days). Relative dose intensity (%) is the ratio of absolute dose intensity divided by the intended dose intensity. In those cases where the relative dose intensity is over 100% due to permitted dose anticipation (i.e. patients receiving more dose than planned), this ratio will be adjusted to 100%.

The options "Dose Reduced" and "Dose Delayed" available in the Treatment Modification item on the treatment exposure CRF pages will be used to calculate delays and dose reductions, respectively. For cycles considered as delayed by the Investigator, the length of the delay will be calculated as:

Duration of cycle delay: Date of the current drug administration – Date of the previous drug administration – the predefined cycle length (i.e., 21 days).

For itraconazole, the percentage of compliance will be calculated by dividing the actual total dose by the intended dose.

If the number of delays or dose reductions are very low, tables will not be presented and only listings will be shown.

#### 7.5 Subsequent Therapies

A listing of the first subsequent therapies received after treatment discontinuation will be shown by study part and treatment sequence group.

## 7.6 Imputation in Incomplete Dates

Dates of certain historical or current clinical activities are key component for statistical analysis. An incomplete date results from a missing day, month or year; in that case, the missing figure can be imputed allowing for the calculation of variables, such duration and time to certain event. However, when all of them, day, month and year, are missing no imputation will be done.

Before randomization/treatment start date

All variables needed to summarize for example prior information (e.g. first diagnosis date) where partial information is available will be subject of imputation by means of SAS programming. If the day of a date is unknown then the imputed day will be 1, if the month is also unknown then the imputed date will 1/July. This assumption will be valid if the imputed date is earlier than the randomization date; otherwise, the imputed date will be the first day of the month of the randomization date (i.e. 01/Randomization month date/year).

#### Between treatment start and end of treatment

All date variables during treatment where information is needed and is not fully available, for example adverse events or concomitant medications, will be subject of imputation by means of SAS programming. If the day of a date is unknown then the imputed day will be 1, if the month and/or year is also unknown then the imputed date will 1/January (this assumption will be valid if the imputed date is not earlier than the treatment start date; otherwise, the imputed date will be the treatment start date).

#### After end of treatment

A conservative approach for the variables collecting information after end of treatment where partial information is available (e.g., follow-up AEs) will be imputed by means of SAS programming. The following rules will be implemented: if the day of a date is unknown then the imputed day will be 1; if the month is also unknown, then the imputed date will be 1/July. This assumption will be valid if the imputed date occurs later than the last drug administration date; otherwise, the imputed date will be the last drug administration date plus 1 day.

#### 7.7 Variable Unit Standardization

Variables reported with different units will be homogenized to standardized variables following the International System of Units (e.g. laboratory tests, biometrical assessments...) unless otherwise specified in the following sections.

## 7.8 Decimal Places, Missing Values and Allowed Assessment Windows

By default, all results will be rounded to one decimal place, except when variables are integer, which will be reported without decimals (e.g., age in years, number of sites, etc.). For representing p-values four decimals will be selected as default but they could be rounded to fewer decimals if necessary.

Missing values will not be imputed. Assessment windows as specified in the clinical protocol will be respected.

#### 7.9 Subgroup Analyses

Safety analysis will be done by study part and sequence treatment arm.

No other subgroup analysis is planned.

## 7.10 Pharmacogenetic Analysis

The analysis of pharmacogenetic data will be detailed and reported in a separate document.

## 7.11 Identification of Fixed or Random Effects Models

Not applicable.

## 7.12 Data Analysis Conventions

All data analysis conventions, data calculations and grouping needed to perform the statistical analysis not included in this SAP will be described in separate document.

## 8 STATISTICAL SOFTWARE

Medidata Rave® EDC will be used for data entry and clinical data management.

Medidata Rave® RTSM will be used for permuted block randomization design and management.

SAS® v.9.4 or superior will be used for all statistical analysis outputs.

## 9 REFERENCES

- 1. Food and Drug Administration (FDA).2001. Guidance for Industry. Statistical approaches to establishing bioequivalence.
- 2. SAS OnlineDoc.

#### 10 APPENDIX I: PATIENTS DISPOSITION

#### 10.1 General Characteristics

The general characteristics analysis will be carried out on the enrolled population.

## 10.1.1 Patient Disposition

The main characteristics of the enrolled patients (inclusion in the study, withdrawal from the study and protocol deviations) will be displayed in this section.

Table 10.1.1.1 Patient accrual by institution

| Part A | | | Part B | | | Part | A+B | _ | |
|--------|-----|------|--------|------|-----|------|-----|----|------|
| S1 ( | TR) | S1 ( | TR) | S2 ( | RT) | S1 ( | TR) | To | otal |
| N | % | N | % | N | % | N | % | N | % |

Institution 1

Institution 2

Total

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.1.1.2 Disposition of patients

Relevant study dates

Date of first consent

Date of first dose/first patient

Date of last consent

Date of first dose/last patient

Date of last dose

Date of last follow up\*

Table 10.1.1.3 Number of patients evaluable for analysis

| Par | t A | | Pa | rt B | | Part | A+B | | |
|------|-----|------|-----|------|-----|------|-----|----|------|
| S1 ( | TR) | S1 ( | TR) | S2 ( | RT) | S1 ( | TR) | To | otal |
| N | % | N | % | N | % | N | % | N | % |

Included

Evaluable for PK

Evaluable for Safety

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

<sup>(\*)</sup> Last follow up date, examination date or procedure before study closure.

| Listing | 10.1 | 1 / Man | -evaluable | nationta |
|---------|-------|---------|------------|----------|
| Lisung | 10.1. | 1.4 Non | -evaruante | batients |

| Not Evaluable for | Study Part | Sequence | Subject | Max. Cycle received | Reason(s) |
|---|---|---|---|---|---|
| PK | | | | | |
| Safety | | | | | |
| ••• | | | | | |

#### 10.1.2 Treatment Discontinuations

#### Table 10.1.2.1 Treatment discontinuation

| Par | t A | | Pa | rt B | | Part | A+B | _ | |
|------|-----|------|------|------|-----|------|-----|----|------|
| S1 ( | TR) | S1 ( | (TR) | S2 ( | RT) | S1 ( | TR) | То | otal |
| N | % | N | % | N | % | N | % | N | % |

Protocol Treatment Completed

Patient moved to

Compassionate Use

Progressive disease

Adverse Events

Patient refusal to treatment

Investigator's decision

Death

Other

Total

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 10.1.2.2 Treatment discontinuation due to related<sup>†</sup> Adverse Events

| Study Part Sequence Tre | atment Subject | Cycle | AE | Preferred | Grade | Relationshi | Serious |
|---|---|---|---|---|---|---|---|
| G <sub>1</sub> | roup* | | reported | term | | p | Event |

Notes: † Related or unknown relationship.

Listing 10.1.2.3 Treatment discontinuation due to non-related Adverse Events

| Study Part Sequence Treatment | Subject | Cycle | AE | Preferred | Grade | Relationshi | Serious |
|---|---|---|---|---|---|---|---|
| Group* | | | reported | term | | p | Event |

<sup>\*</sup> ITZ+LRB / LRB

Listing 10.1.2.4 Reasons for treatment discontinuation other than Progressive Disease

| Study | Part | Sequence | Subject | Max. Cycle received | Reason | Specify |
|-------|------|----------|---------|---------------------|--------|---------|

<sup>\*</sup> ITZ+LRB / LRB

Table 10.1.2.5 Reasons for study discontinuation

| Total S1 (TR) S1 (TR) S2 (RT) S1 (TR) N % N % N % N % N % | Par | t A | | Par | rt B | | Part . | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 ( | TR) | S1 ( | TR) | S2.( | RT) | S1 ( | TR) | То | tal |
| | | % | , | % | | % | | % | N | % |

Patient's follow-up completed

Patient moved to

Compassionate Use

Study termination

(clinical cut-off)

Withdrawal of consent

Death

Never treated

Lost to follow up

Other

Total

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 10.1.2.6 Reasons for treatment discontinuation due to other reason

| Study Part | Sequence | Subject | Max. Cycle received | Other, specify |
|------------|----------|---------|---------------------|----------------|

Listing 10.1.2.7 Patients never treated

| Study Part | Sequence | Subject | Reason |
|------------|----------|---------|--------|
| | | - | |

#### 10.1.3 **Protocol Deviations**

Listing 10.1.3.1 Relevant protocol deviations

| Study Part | Sequence | Subject | Cycle | Protocol deviation Specify Deviation |
|---|---|---|---|---|
| | | | | Туре |

Notes: See 16.2.2 for a full listing (relevant and non-relevant).

#### 10.2 Patient Characteristics

Baseline/screening characteristics of all enrolled patients (enrolled population) will be described.

#### 10.2.1 Demographic and Other Baseline Characteristics

Table 10.2.1.1 Patients characteristics at baseline: Gender

| Par | t A | | Pa | rt B | | Part . | A+B | | |
|------|-----------------|---|------|------|------|---------|-----|------|---|
| S1 ( | S1 (TR) S1 (TR) | | S2 ( | (RT) | S1 ( | S1 (TR) | | otal | |
| N | % | N | % | N | % | N | % | N | % |

Gender

Male

Female

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.1.2 Patients characteristics at baseline: Race

| Part . | A | | Par | t B | | Part . | A+B | | |
|---|---|---|---|---|---|---|---|---|---|
| S1 (TR) S1 (TR) | | S2 (RT) S1 (T | | | To T | | otal | | |
| <br>N | % | N | % | N | % | N | % | N | % |

Race

White

Black Asian

- ---

Other (Specify)

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.1.3 Patients characteristics at baseline: Age

| _ | Part A | Par | t B | Part A+B | _ |
|---|---------|---------|---------|----------|-------|
| _ | | | | | Total |
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | |

Age at entry (years)

N

Median (range)

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 10.2.1.4 Patients characteristics at baseline: Pregnancy Test

| | Par | Part A | | Part B | | | Part A+B | | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 ( | S1 (TR) | | S1 (TR) S2 (RT) | | (RT) | S1 (TR) | | Total | |
| | N | % | N | % | N | % | N | % | N | % |
| Pregnancy Test | | | | | | | | | | |

| | Pai | t A | | Pa | rt B | | Part | A+B | _ | |
|----------|------|-----|------|-----|------|------|------|-----|----|------|
| | S1 ( | TR) | S1 ( | TR) | S2 ( | (RT) | S1 ( | TR) | To | otal |
| | N | % | N | % | N | % | N | % | N | % |
| Positive | 11 | | | | | | | | | - |

Positive

Negative

NA (Specify)

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.1.5 Patients characteristics at baseline: Adequate contraception

| _ | Par | t A | | Part B | | | Part | A+B | _ | |
|---|------|-----|------|--------|------|------|------|-----|----|------|
| | S1 ( | TR) | S1 ( | (TR) | S2 ( | (RT) | S1 ( | TR) | To | otal |
| _ | N | % | N | % | N | % | N | % | N | % |

Adequate

contraception

Yes

No

NA (Specify)

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

## 10.2.2 Medical History

Listing 10.2.2.1 Ongoing medical history

| Study Part | Sequence | Subject | Description | Onset date |
|------------|----------|---------|-------------|------------|

## 10.2.3 Cancer History

Table 10.2.3.1 First diagnosis: Tumor type and stage at diagnosis

| Par | t A | | Pa | rt B | | Part | A+B | _ | |
|------|-----|------|------|------|-----|------|-----|----|------|
| S1 ( | TR) | S1 ( | (TR) | S2 ( | RT) | S1 ( | TR) | To | otal |
| N | % | N | % | N | % | N | % | N | % |

Tumor Type

Lung

Kidney

Prostate cancer

Stage at Diagnosis

Early

Locally advanced

Metastatic

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.3.2 First diagnosis: Time from first diagnosis to first infusion

| | Part A | Part A Part B | | Part A+B | _ |
|---|---|---|---|---|---|
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | Total |
| Time form first diagnosis to first | | | | | |
| infusion (years) †<br>N | | | | | |
| Median (range) | | | | | |

<sup>&</sup>lt;sup>†</sup> Time from first diagnosis to first infusion: defined as the date of first infusion minus date of first diagnosis.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.3.3 Current disease: Time from last PD to first infusion

| | Part A | Par | rt B | Part A+B | _ |
|---|---|---|---|---|---|
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | Total |
| Time from last PD <sup>†</sup> to first | | | | | 11 11 |

Time from last PD<sup>†</sup> to firs infusion (months)<sup>‡</sup>

N

Median (range)

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.3.4 Current disease: Sites of disease involvement

| _ | Part | A | | Par | t B | | Part A | A+B | _ | |
|---|-------|----|------|-----|------|-----|--------|-----|----|------|
| | S1 (T | R) | S1 ( | TR) | S2 ( | RT) | S1 ( | TR) | To | otal |
| _ | N N | % | N | % | | % | | % | N | % |

Site of disease

involvement

Lung

Liver

Lymph node

• • •

Other (Specify)

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 10.2.3.5 No. of sites of disease involvement

| | Par | t A | | Pa | rt B | | Part | A+B | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 ( | S1 (TR) | | S1 (TR) | | S2 (RT) | | S1 (TR) | | otal |
| | N | % | N | % | N | % | N | % | N | % |
| 1 | | | | | | | | | | |

<sup>†</sup> Last PD will be taken from the Cancer history form.

<sup>&</sup>lt;sup>‡</sup> Time from last PD to first infusion: date first infusion minus date of last progression before study entry.

| | P | art A | | Pa | rt B | | Part | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 | S1 (TR) | | S1 (TR) | | S2 (RT) | | S1 (TR) | | otal |
| | N | % | N | % | N | % | N | % | N | % |
| <br>≥ N sites<br>Total | | | | | | | | | | |
| Total | | | | | | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.3.6 Summary statistics: No. of sites of disease involvement

| | Part A | Pa | rt B | Part A+B | _ |
|---------------------|---------|---------|---------|----------|-------|
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | Total |
| N<br>Median (range) | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

## 10.2.4 Previous Anticancer Therapy Summary

Table 10.2.4.1 Prior surgery

| Par | t A | Pa | rt B | | Part | A+B | _ | |
|------|---------|---------|------|---------|------|---------|---|------|
| S1 ( | S1 (TR) | S1 (TR) | | S2 (RT) | | S1 (TR) | | otal |
| N | | % | N | % | N | % | N | % |

Prior surgery

Yes

No

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.2 Prior radiotherapy

| | Par | t A | | Par | rt B | | Part | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 ( | S1 (TR) | | S1 (TR) | | S2 (RT) | | TR) | To | otal |
| <del>-</del> | N | % | N % | | N % | | N % | | N | % |

Prior radiotherapy

Yes

No

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.3 Prior anticancer medical therapy for study disease: Setting

| Par | t A | Pa | rt B | | Part | A+B | _ | |
|------|---------|---------|------|------|---------|-----|----|------|
| S1 ( | S1 (TR) | S1 (TR) | | (RT) | S1 (TR) | | To | otal |
| N | | % | N | % | N | % | N | % |

Setting

Neoadjuvant

Adjuvant

Advanced

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.4 Prior anticancer medical therapy for study disease: No. of prior lines

| Par | t A | | Pa | rt B | | Part | _ | | |
|------|---------|---|---------|------|------|---------|---|----|------|
| S1 ( | S1 (TR) | | S1 (TR) | | (RT) | S1 (TR) | | To | otal |
| N | % | N | % | N | % | N | % | N | % |

No. of prior lines

1 line

2 lines

3 lines

>= 4 lines

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.5 Prior anticancer medical therapy for study disease: Summary of prior lines

| | | _ | Part A | Par | t B | Part A+B | _ |
|---------|-----------|-------|---------|---------|---------|----------|-------|
| | | | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | Total |
| No. | of | prior | () | 21 (11) | () | 22 (22) | |
| chemoth | erapy lin | es | | | | | |
| N | | | | | | | |
| Median | (range) | | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.6 Prior anticancer medical therapy for study disease: Best response to last therapy

| | Par | t A | | Pa | rt B | | Part | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| Best response to last prior | S1 ( | Part A | | S1 (TR) | | S2 (RT) | | TR) | To | otal |
| therapy | N | % | N | % | N | % | N | % | N | % |
| | 1/ | 70 | 1/ | 70 | 1/ | 70 | 1/ | 70 | 1/ | 70 |

Complete Response Partial Response Stable Disease Progressive Disease Not Evaluable Unknown Not Applicable

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.7 Prior anticancer medical therapy for study disease: Time to progression of last therapy

| _ | Part A | Par | rt B | Part A+B | _ |
|---|---|---|---|---|---|
| Time to progression (months) | | | | | Total |
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | |
| N | | | | | |
| Median (range) | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

## 10.2.5 Physical Examination, ECOG, Vital Signs, LVEF and ECG

Table 10.2.5.1 Physical examination at baseline

| | Par | t A | | Par | rt B | | Part | A+B | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Physical examination | S1 ( | S1 (TR) | | S1 (TR) | | S2 (RT) | | S1 (TR) | | otal |
| | N | % | N | % | N | % | N | % | N | % |
| Normal<br>Abnormal | | | | | | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 10.2.5.2 Physical examination at baseline: abnormalities

| Study Part | Sequence | Subject | Description |
|------------|----------|---------|-------------|

Table 10.2.5.3 Weight, height and BSA at baseline

| | Part A | Par | rt B | Part A+B | _ |
|---------------------|---------|---------|---------|----------|-------|
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | Total |
| | | | , , | , , , | |
| Weight (kg) | 11 | | | | |
| N<br>Median (range) | | | | | |
| Height (cm) | | | | | |

Median (range)

BSA (m<sup>2</sup>)

N

Median (range)

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.5.4 ECOG Performance Status at baseline

| | Pai | t A | | Par | rt B | | Part | A+B | -<br>Tr. 4 1 | |
|---|---|---|---|---|---|---|---|---|---|---|
| ECOG | S1 ( | S1 (TR) | | S1 (TR) | | S2 (RT) | | S1 (TR) | | Total |
| | N | % | N | % | N | % | N | % | N | % |
| 0 | | | | | | | | | | |
| 1 | | | | | | | | | | |
| ••• | | | | | | | | | | |
| Total | | | | | | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 10.2.5.5 Vital signs at baseline

| | Part A | Par | rt B | Part A+B | <u> </u> |
|---|---|---|---|---|---|
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | Total |
| Heart rate (Beats/minute) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Temperature (°C) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Blood pressure systolic (mmHg) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Blood pressure diastolic (mmHg) | | | | | |

| | Part A | Pa | rt B | Part A+B | |
|----------------|---------|---------|---------|----------|-------|
| | | | | | Total |
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | |
| N | | | | | |
| Madian (ranga) | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.5.6 ECG<sup>†</sup> pre infusion at baseline

| | Pai | t A | | Par | t B | | Part A | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 ( | S1 (TR) | | S1 (TR) S2 (RT) | | | S1 (TR) | | To | otal |
| | N | % | N | % | N | % | N | % | N | % |
| Result<br>Normal | '' | | | | | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

† Worst result of the three ECGs replicates will be used as baseline value.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.5.7 ECG<sup>†</sup> pre infusion at baseline

| | Par | t A | | Par | rt B | | Part . | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 ( | TR) | S1 ( | (TR) | S2 ( | (RT) | S1 ( | TR) | То | otal |
| | N | % | N | % | N | % | N | % | N | % |
| PR interval (msec) | | | | | | | | | | |
| N | | | | | | | | | | |
| Median (range) | | | | | | | | | | |
| Heart rate (bpm) | | | | | | | | | | |
| N | | | | | | | | | | |
| Median (range) | | | | | | | | | | |
| QT interval (msec) | | | | | | | | | | |
| N | | | | | | | | | | |
| Median (range) | | | | | | | | | | |
| Bazett's corrected QT | | | | | - | | | | | |
| N | | | | | | | | | | |
| Median (range) | | | | | | | | | | |
| N D | 1 ( | • | 1 , 1 | , 1 | | 1 | 1' 11 | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

† Mean of the three ECGs replicates will be used as a baseline value.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

| T | isting | 10.2 | 5.8 | Patients | with | ahnormal | ا ا | ectrocardiogram |
|---|---|---|---|---|---|---|---|---|
| | лышш | 10.2 | | T allellis | willi | aunoma | | CCHOCAIGIOPIAIII |

| Study Part | Sequence | Subject | ECG no. | Abnormality | PR interval (msec) | <br>` | |
|---|---|---|---|---|---|---|---|
| | | | | | | | QT |

#### Table 10.2.5.9 LVEF at baseline

| | Par | t A | | Pa | rt B | | Part | A+B | _ | |
|---|------|-----|------|------|------|------|------|-----|----|------|
| | S1 ( | TR) | S1 ( | (TR) | S2 ( | (RT) | S1 ( | TR) | То | otal |
| • | N | % | N | % | N | % | N | % | N | 9/ |

Result Normal Abnormal

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 10.2.5.10 Patients with abnormal LVEF

| Study Part | Sequence | Subject | Result | Method | Value (%) | Lower limit (%) | Abnormalities |
|---|---|---|---|---|---|---|---|

Notes: Significant and non-significant abnormalities

#### Table 10.2.5.11 LVEF value at baseline

| | Par | t A | | Par | rt B | | Part | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| LVEF (%) | S1 (TR) | | S1 (TR) | | S2 (RT) | | S1 (TR) | | Total | |
| | N | % | N | % | N | % | N | % | N | % |
| MUGA | | 11 | 11 | | | | | ** | | |
| N | | | | | | | | | | |
| Median (range) | | | | | | | | | | |
| ЕСНО | | | | | | | | | | |
| N | | | | | | | | | | |
| Median (range) | | | | | | | | | | |
| Both | | | | | | | | | | |
| N | | | | | | | | | | |
| Median (range) | | | | | | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

# 10.2.6 Hematological Evaluation at Baseline

Table 10.2.6.1 Hematology abnormalities at baseline<sup>†</sup>

| | P | art A | | | Part B | | | Part A+ | -В | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Si | 1 (TR) | S | S1 (TR) | | S2 (RT) | | S1 (TF | 2) | Tot | al |
| All grades | Gr 1 | * | All<br>grades | Gr 1 | * | All<br>grades | Gr 1 | * | All<br>grades | Gr 1 | * |
| N % | N % | N % | N % | N % | N % | N % | N % | N % | N % | N % | N % |

Anemia Leukopenia Lymphopenia Neutropenia Thrombocytopenia

Defined as the last value recorded before or on the date of first infusion.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test. \* Gr 1, Gr 2, Gr 3, Gr 4

Table 10.2.6.2 Median and range for hematology parameters at baseline<sup>†</sup>

| | | Pa | art A | P | art B | ] | Part A+B | |
|---|---|---|---|---|---|---|---|---|
| | | S1 | (TR) | S1 (TR) | S2 (F | RT) | S1 (TR) | Total |
| Hemoglobin | (g/dL) | | | | * | | | |
| N | , | | | | | | | |
| Median (ran | ge) | | | | | | | |
| WBC (10%L) | ) | | | | | | | |
| N | | | | | | | | |
| Median (ran | ge) | | | | | | | |
| Lymphocyte | s (10%L) | | | | | | | |
| N | | | | | | | | |
| Median (ran | ge) | | | | | | | |
| N | | | | | | | | |
| Median (ran | ge) | | | | | | | |
| | | | | date of first inf | | | | |
| | | | | juence assigned | | | | |
| S1, Sequence | e 1; S2, Seque | nce 2; TR, to | est-reference | ; RT, reference | -test. | | | |
| Listing 10.2 | 2.6.3 Hemato | logical abr | normalities | at baseline (gr | rade $\geq 2$ ) | | | |
| Study Part | Sequence | Subject | Lab. Test | Examination date | Value | Std. Value | Std. Unit | Grade |
| | | | | | | | - | |
| | - | | - | | | | - | |

Listing 10.2.6.4 Hematological tests not assessed at baseline

| Study Part | Sequence | Subject | Lab. Test |
|------------|----------|---------|-----------|

## 10.2.7 Biochemical Evaluation at Baseline

Table 10.2.7.1 Biochemical abnormalities at baseline<sup>†</sup>

| | P | art A | | | Part B | | Part A+B | |
|---|---|---|---|---|---|---|---|---|
| | Si | (TR) | S | S1 (TR) | S2 (R' | Т) | S1 (TR) | Total |
| All grades | Gr 1 | ** | All<br>grades | Gr 1 | ** All grade | es Gr 1 | | All Gr 1** |
| N % | N % | N % | N % | N % | N % N 9 | % N % | N % N | % N % N % |

ALT increased AST increased

Defined as the last value recorded before or on the date of first infusion.

<sup>\*</sup>Creatinine increased, hyperglycemia, hypoglycemia, CPK increased, GGT increased, bilirubin increased, hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, hypercalcemia, hypocalcemia.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>\*\*</sup> Gr 1, Gr 2, Gr 3, Gr 4

Table 10.2.7.2 Median and range for biochemical parameters at baseline<sup>†</sup>

| | | Part A | | Part B | | Part A+B | |
|---|---|---|---|---|---|---|---|
| | | S1 (TR) | S1 ( | (TR) S | 2 (RT) | S1 (TR) | Total |
| ALT (xULN) | | | | | | | |
| N | | | | | | | |
| Median (range | e) | | | | | | |
| AST (xULN) | | | | | | | |
| N | | | | | | | |
| Median (range | e) | | | | | | |
| N | | | | | | | |
| Median (range | | | | | | | |
| Defined as the | last value reco | rded before or | on the date of | first infusion. | | | |
| art A, patients | s assigned to Se | equence 1; Part | B, sequence | assigned random | ly. | | |
| · • | l; S2, Sequence | | | C | 3 | | |
| Listing 10.2.7 Study Part | 7.3 Biochemic<br>Sequence | al abnormali<br>Subject | ies at baseli<br>Lab. Test | ne (grade ≥ 2) Examination date | Value | Std. Value | Grade |
| | | , | | - Cutt | | | |
| | | | | | | <del></del> | |
| | | al abnormali | ties not asses | sed at baseline | | | |
| Listing 10.2.7<br>Study | | al abnormali<br>Sequ | | sed at baseline<br>Subj | | Lab. 7 | Γest |
| | | | | | | Lab. 7 | Γest |

## 10.2.8 Coagulation Evaluation at Baseline

Table 10.2.8.1 Coagulation abnormalities at baseline<sup>†</sup>

| | Part A | | | Part B | | Part A+B | |
|---|---|---|---|---|---|---|---|
| | S1 (TR) | | S1 (TR) | S | 2 (RT) | S1 (TR) | Total |
| All<br>grades Gr | 1* | All<br>grades | Gr 1 | * g | All Gr 1 | * All grades | Gr 1* |
| N % N | % N % | N % | N % | N % N | N % N % | N % N % | N % N% |

#### INR increased

Defined as the last value recorded before or on the date of first infusion.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Listing 10.2.8.2 INR increased at baseline (grade  $\geq$  2)

| Study Part Sequ | uence Subject | Lab. Test | Examination date | Value | Std. Value | Grade |
|---|---|---|---|---|---|---|

<sup>\*</sup>Gr 1, Gr 2, Gr 3, Gr 4

Listing 10.2.8.3 INR not assessed at baseline

| Study Part | Sequence | Subject | Lab. Test |
|------------|----------|---------|-----------|

## 10.2.9 Signs and Symptoms at Baseline

Signs and symptoms refer to any AE with onset date before the first treatment dose.

Table 10.2.9.1 Signs and symptoms at baseline (MedDRA coded)

| | Par | t A | | Par | rt B | | Part | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA SOC/PT <sup>†</sup> | S1 ( | TR) | S1 ( | (TR) | S2 ( | (RT) | S1 ( | TR) | То | otal |
| | N | % | N | % | N | % | N | % | N | % |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

†SOC: System Organ Class; PT: Preferred Term

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.9.2 Signs and symptoms at baseline

| | Part A | | | Part B | | | | Part A+B | | |
|---|---|---|---|---|---|---|---|---|---|---|
| No. of signs and symptoms per patient – | S1 (TR) | | S1 ( | S1 (TR) | | S2 (RT) | | S1 (TR) | | otal |
| | N | % | N | % | N | % | N | % | N | % |
| 0 | | | | | | | | | | |
| 1 2 | | | | | | | | | | |
| ≥ 3 | | | | | | | | | | |
| Total | • | - | | | | • | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.9.3 Summary of signs and symptoms at baseline

| N C' 1 | Part A Part B | | t B | Part A+B | |
|---|---|---|---|---|---|
| No. of signs and symptoms per patient | | | | | Total |
| per patient | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | |
| N | | | | | |
| Median (range) | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Listing 10.2.9.4 Signs and symptoms at baseline (grade  $\geq 2$ )

| Study Part | Sequence | Subject | Sign/symptom | MedDRA<br>Preferred<br>Term | Grade | Onset date | Relationship |
|---|---|---|---|---|---|---|---|

## 10.2.10 Concomitant Medication at Baseline

Concomitant medication at baseline according to the ATC classification.

Table 10.2.10.1 Concomitant medication at baseline (ATC levels1, 2 and 4)

| | Pai | t A | | Pa | rt B | | Part | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| Concomitant medication | S1 ( | (TR) | S1 (TR) | | S2 (RT) | | S1 (TR) | | Total | |
| | N | % | N | % | N | % | N | % | N | % |

Alimentary tract and metabolism

Antacids

Magnesium compounds Magnesium adipate

. . .

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

#### 11 APPENDIX II: SAFETY ANALYSIS

#### 11.1 Extent of Exposure

This analysis will be carried out on evaluable patients for the safety population.

#### 11.1.1 Treatment Administration

Table 11.1.1.1 Number of cycles administered<sup>†</sup>

| Par | t A | | Pai | t B | | Part . | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|
| S1 (TR) S1 (TF | | TR) | R) S2 (RT) | | S1 (TR) | | Total | | |
| N | % | N | % | N | % | N | % | N | % |
| | S1 ( | S1 (TR) | S1 (TR) S1 ( | S1 (TR) S1 (TR) | S1 (TR) S1 (TR) S2 ( | S1 (TR) S1 (TR) S2 (RT) | S1 (TR) S1 (TR) S2 (RT) S1 ( | S1 (TR) S1 (TR) S2 (RT) S1 (TR) | S1 (TR) S1 (TR) S2 (RT) S1 (TR) |

<sup>1</sup> cycle

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Table 11.1.1.2 Summary of number of cycles administered<sup>†</sup> and time on treatment

| | Part A | Part B | | Part A+B | _ |
|----------------------------|---------|---------|---------|----------|-------|
| | | | | | Total |
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | |
| No. of cycles administered | | | | | |
| per patient | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Time on treatment (weeks)* | | | | | |
| N | | | | | |
| Median (range) | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 11.1.1.3 Dose information by study part and sequence

| _ | Part A | Part B | | Part A+B | _ |
|---|---|---|---|---|---|
| | | | | | Total |
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | |
| | | | Lurbinectedin | | |
| Cumulative dose (mg/m <sup>2</sup> ) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Dose intensity (mg/m²/week) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Relative dose intensity (%) | | | | | |
| N | | | | | |
| Median (range) | | | | | |

<sup>2</sup> cycles

<sup>3</sup> cycles

<sup>†</sup> Including when lurbinectedin is administered both alone and in combination with itraconazole.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†</sup> Including when lurbinectedin is administered both alone and in combination with itraconazole.

<sup>\*</sup>Time on treatment is defined as the last administration date of lurbinectedin plus 31 days, death or the start date of the new therapy, whichever comes first, minus the first administration date of lurbinectedin.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.
| | Part A | Par | t B | Part A+B | _ |
|----------------------|---------|---------|--------------|----------|-------|
| | | | | | Total |
| | S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | |
| | | | Itraconazole | | |
| Cumulative dose (mg) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Compliance (%) | | | | | |
| N | | | | | |
| Median (range) | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

## 11.1.2 Cycle Delays

Table 11.1.2.1 Summary of lurbinectedin dose delays

| - | Pai | t A | | Par | t B | | Part | A+B | | _ |
|---|---|---|---|---|---|---|---|---|---|---|
| _ | S1 ( | (TR) | S1 | (TR) | S2 ( | RT) | S1 ( | TR) | Т | otal |
| | N | % | N | % | N | % | N | % | N | % |
| No. of patients treated | | | | | × | | | | | - |
| No. of patients susceptible to have dose delay † | | | | | | | | | | |
| No. of patients with any do | se | | | | | | 1.1 | | | |
| delay | | | | | | | | | | |
| Drug related <sup>‡</sup> AE | | | | | | | | | | |
| Non-drug related AE | | | | | | | | | | |
| Other reason | | | | | | | | | | |
| No. of cycles administered | | | | | | | | | | |
| No. of cycles susceptible to have dose delay †† | ve | | | | | | | | | |
| No. of cycles with any dose delay | ,;# | | | | : | | | | | |
| Drug related <sup>‡</sup> AE | y · · | | | | | | | | | |
| Non-drug related AE | | | | | | | | | | |
| Other reason | | | | | | | | | | |
| † Excluding patients who receive | od oply t | ha first ar | ro10 | | | | | | | |

Excluding patients who received only the first cycle.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.1.2.2 Length of delay

| | Par | t A | | Pa | rt B | | Part | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 ( | TR) | S1 ( | (TR) | S2 ( | (RT) | S1 ( | TR) | То | otal |
| | N | % | N | % | N | % | N | % | N | % |
| Length of delay <sup>‡‡</sup> | | | | | | | | | | |
| ≤ 2 days | | | | | | | | | | |
| ≤ 7 days | | | | | | | | | | |
| $> 7$ to $\le 14$ days | | | | | | | | | _ | |

<sup>‡</sup> Related or unknown relationship

<sup>††</sup> All cycles excluding first cycle

<sup>‡‡</sup> Denominator = Number of cycles susceptible to have dose delay

†‡ Denominator = Number of cycles susceptible to have dose delay

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.1.2.3 Dose delays

| Study Part Sequence Treatment Group* | Subject | Cycle | Delay (days) | Reason for delay |
|---|---|---|---|---|

<sup>\*</sup> ITZ+LRB / LRB

#### 11.1.3 Dose Reductions

Table 11.1.3.1 Summary of lurbinectedin dose reductions

| | D | -4 A | | n | 4 D | | D4 | A + D | | |
|---|---|---|---|---|---|---|---|---|---|---|
| - | Pai | t A | | Pai | t B | | Part . | A+B | - <sub>T</sub> | . 1 |
| - | S1 ( | (TR) | S1 ( | (TR) | S2 ( | RT) | S1 ( | TR) | 10 | otal |
| | N | % | N | % | N | % | N | % | N | % |
| No. of patients treated | | | | | | | | | | |
| No. of patients susceptible to have dose reduction † No. of patients with any do reduction | se | | | | | | | | | |
| Drug related <sup>‡</sup> AE Non-drug related AE | | | | | | | | | | |
| Other reason | | | | | | | | | | |
| No. of cycles administered | | ************************************** | 11 | | : | | ·· | | | |
| No. of cycles susceptible to hadose reduction † | ve | | | | | | | | | |
| No. of cycles with any do reduction <sup>#</sup> Drug related <sup>‡</sup> AE Non-drug related AE | se | | | | | | | | | |

<sup>†</sup> Excluding patients who received only the first cycle.

Other reason

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.1.3.2 Dose reductions

| Study Part | Sequence | Treatment Subject<br>Group* | Cycle | Lurbinectedin intended dose (mg/m²) | Reason for dose Specify reduction |
|---|---|---|---|---|---|

<sup>\*</sup> ITZ+LRB / LRB

<sup>‡</sup> Related or unknown relationship

<sup>††</sup> All cycles excluding first cycle

<sup>‡‡</sup> Denominator = Number of cycles susceptible to have dose delay/reduction

# 11.1.4 Any Other Dose Modifications

Listing 11.1.4.1 Dose interruptions for lurbinectedin

| Study Part | Sequence | Treatment Group* | Subject | Cycle | Date | Reason for interruption | Specify |
|---|---|---|---|---|---|---|---|
| * ITZ+LRB / I | LRB | · | | | | | |

# Listing 11.1.4.2 Dose Omissions for lurbinectedin

| Group* | | Date | Cycle | Subject | Treatment | Sequence | Study Part |
|---|---|---|---|---|---|---|---|
| Group | omission | | | | Group* | | |

<sup>\*</sup> ITZ+LRB / LRB

Listing 11.1.4.3 Dose not taken according to protocol for Itraconazole

| Study Part | Sequence | Treatment<br>Group* | Subject | Cycle | Date | Reason for omission | Specify |
|---|---|---|---|---|---|---|---|

<sup>\*</sup> ITZ+LRB / LRB

#### 11.2 Adverse Events (AEs)

This analysis will be carried out on evaluable patients for the safety population.

All adverse events tables will be listed by study part and sequence and differentiating by treatment (Test, Reference or both). Additional groups could be done (such as PM01183 alone or in combination) if required, and a sequential number will be added at the end of the table number.

AEs consisting of laboratory abnormalities (e.g., neutropenia) may be under-reported as AEs. Since these events are better evaluated using objective laboratory results, laboratory abnormalities will be discussed in Section 11.4.

The type of toxicity and worst grade or severity by cycle and by patient will be summarized according to System Organ Class (SOC) and Preferred Term (PT) as per the MedDRA dictionary. Subsequent grouping of similar or clinically related items might be appropriate at the time of the analysis. Tables will be organized by category of events using SOC and PT. Grades could be presented by separate or any other grouping at the time of the analysis.

## 11.2.1 Display of Adverse Events

Table 11.2.1.1 Summary of adverse events

| Par | rt A | | Pai | rt B | |
|------|------|------|------|------|------|
| S | 1 | S | 1 | S | 32 |
| Т | R | Т | R | R | T |
| N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

No. of patients with any AE

No. of patients with any treatment-related AE

Patients with any grade 3/4 AE

Patients with any grade 4 AE

No. of patients with any grade 3/4 treatment-related<sup>†</sup> AE

No. of patients with any grade 4 treatment-related  $^{\dagger}$  AE

No. of patients with any SAE

No. of patients with any treatment-related SAE

No. of patients with any grade 3/4 SAE

No. of patients with any grade 4 SAE

Any grade 3/4 treatment-related<sup>†</sup> SAE

Any grade 4 treatment-related† SAE

No. of patients with deaths associated with AEs

No. of patients with deaths associated with treatment-related<sup>†</sup>

AEs

No. of patients with dose delays associated with AEs

No. of patients with dose delays associated with treatment-

related<sup>†</sup> AEs

No. of patients with dose reductions associated with AEs

No. of patients with dose reductions associated with

treatment-related†AEs

No. of patients with dose interruptions associated with AEs

No. of patients with dose interruptions associated with

treatment-related† AEs

| Part | A+B | |
|------|------|-------|
| S | 51 | Total |
| Т | R | |
| N(%) | N(%) | N(%) |

No. of patients with any AE

No. of patients with any treatment-related † AE

Patients with any grade 3/4 AE

Patients with any grade 4 AE

No. of patients with any grade 3/4 treatment-related<sup>†</sup> AE

No. of patients with any grade 4 treatment-related<sup>†</sup> AE

No. of patients with any SAE

No. of patients with any treatment-related SAE

No. of patients with any grade 3/4 SAE

No. of patients with any grade 4 SAE

Any grade 3/4 treatment-related<sup>†</sup> SAE

Any grade 4 treatment-related<sup>†</sup> SAE

No. of patients with deaths associated with AEs

No. of patients with deaths associated with treatment-related<sup>†</sup>

AEs

No. of patients with dose delays associated with AEs

No. of patients with dose delays associated with treatment-

related† AEs

No. of patients with dose reductions associated with AEs

No. of patients with dose reductions associated with

treatment-related†AEs

No. of patients with dose interruptions associated with AEs

No. of patients with dose interruptions associated with

treatment-related† AEs

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

† Related to both or lurbinectedin or itraconazole or with unknown relationship.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

Supplementary tables describing the adverse event toxicity grades or laboratory abnormality grades 1,2,3,4,5 and grade 1-5 will be added below the tables with aggregated severity grades show in sections 11.2.1, 11.3.1, 11.4.1 and 11.4.2 as shown in table 11.2.1.2

Table 11.2.1.2 Treatment related† (or with unknown relationship) Adverse Events. Worst grade by treatment

| | | | Pa | art A | | |
|--------|------------|------------|-------|------------|------------|------|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | Gr ≥4 | All grades | $Gr \ge 3$ | Gr≥4 |
| 500/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | | | Pai | rt B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | S | 1 | | | | | S | 52 | | |
| | T | | R | | | | R | | T | | |
| SOC/PT | All grades Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 |
| | N(%) N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| All $Gr \ge 3$ $Gr \ge 4$ All $Gr \ge 3$ $Gr \ge 4$ All grades $Gr \ge 3$ | |
|---|---|
| SOC/PT grades - grades - grades - | Gr≥4 |
| N(%) N(%) N(%) N(%) N(%) N(%) N(%) | N(%) |

| | | | | | | Part | : A | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <del></del> | | - | Γ | | 1 441 | | | I | ₹ | | |
| GO G/PCF | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 |
| SOC/PT | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| | | | | | | Part B | (S1) | | | | | |
| | 11 | | - | Γ | | | | | I | ? | | |
| SOC/PT | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 |
| 30C/F1 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| ••• | | | | | | | | | | | | - |
| | 11 | | | | | Part B | (S2) | | | | | |
| | | | I | ? | | | | | r | Γ | | |
| SOC/PT | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 |
| 50011 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| ••• | | | | - | - | - | | | | - | - | |
| | :: | | | | | Part A+ | B (S1) | | | | | |
| | 11: | | - | Γ | | | | | J | ? | | |
| SOC/PT | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 |
| 550/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Total

| SOC/PT | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 |
|--------|------|------|------|------|------|---------|
| 50011 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 11.2.1.3 Lurbinectedin related† Adverse Events. Worst grade by treatment

| | | | Pa | art A | | |
|--------|------------|------------|--------|------------|------------|--------|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr ≥ 4 |
| 500/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | C | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | <u> </u> | 1 | | | | | S | 2 | | |
| | T | R | | | | R | | T | | |
| All SOC/PT grades | $Gr \ge 3$ $Gr \ge 4$ | All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr ≥ 4 |
| N(%) | N(%) N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | Part A- | +B (S1) | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | T | | | R | | | Total | |
| SOC/PT | All<br>grades | Gr≥3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr ≥ 4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

Table 11.2.1.4 Itraconazole related Adverse Events. Worst grade by treatment

| | | | Pa | art A | | |
|--------|------------|------------|--------|------------|------------|------|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr≥4 |
| 300/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | | | Pai | Part B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | S | 51 | | | | | S | 2 | | |
| | T | | | R | | | R | | T | | |
| SOC/PT | All<br>grades Gr≥ | 3 Gr ≥4 | All grades | $Gr \ge 3$ | Gr ≥4 | All grades | $Gr \ge 3$ | Gr ≥4 | All grades | Gr ≥ 3 | Gr ≥4 |
| | N(%) N(% | (a) N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | Part A- | +B (S1) | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | T | | | R | | | Total | |
| SOC/PT | All grades | Gr ≥ 3 | Gr ≥4 | All grades | Gr≥3 | Gr ≥4 | All grades | $Gr \ge 3$ | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship. Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2. T, Test (ITZ+LRB); R, Reference (LRB alone: NA).

Table 11.2.1.5 Treatment related<sup>†</sup> (or with unknown relationship) Adverse Events. Worst grade per patient

| | | | | | | Part A | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | T | | 1 41 | | | F | ₹ | | |
| COC/DT | All | grades | Gr | ≥ 3 | Gr | ≥ 4 | All g | rades | Gr | ≥ 3 | Gr | <u>≥4</u> |
| SOC/PT | N | V(%) | N | (%) | N( | %) | N( | %) | N( | %) | N( | %) |
| ••• | | | | | - | | | | | | | |
| | | | | | | Par | t B | | | | | |
| | | | 5 | S1 | | | | | S | 2 | | |
| | | T | | | R | | | R | | | T | |
| SOC/PT | All<br>grade | es Gr≥3 | 3 Gr≥4 | All<br>grades | Gr≥3 | Gr≥4 | All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr≥3 | Gr |
| | N(%) | ) N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N( |
| | | | Part A+ | -B (S1) | | | | | т | otal | | |
| | | T | | | R | | | | 1 | Otai | | |
| SOC/PT | All<br>grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 | 4 All | grades | Gı | : ≥ 3 | Gr | ≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | ) N | J(%) | N | (%) | N( | %) |

Notes: Percentage is based on number of patients by study part and sequence, when applicable. A supplementary Table 11.2.1.5supp will be created with grades 1,2,3,4,5.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2. T, Test (ITZ+LRB); R, Reference (LRB alone).

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

Table 11.2.1.6 Lurbinectedin related† Adverse Events. Worst grade per patient

| | | P | Part A | | Part A Part B | | | | | | Part A+B | | | | | _ | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | | | | | | | | | | | | | | | | | , | Total | |
| | | S1 | (TR | ?) | | 5 | S1 (T | TR) | | | S2 ( | RT) | | | S1 | (TR) | ) | | | |
| | All<br>grades | $G_r > 2$ | Gr. | <u> </u> | A | .11 | G: | <u></u> | C۳ | <u> </u> | A | 11 | Gn. | <u> </u> | G: | <u></u> | Al | 1 | Gr≥ | Gr ≥ 4 |
| | grades | Gi ≥ 3 | GI : | < <b>4</b> | gra | des | Gi | ≥ 3 | GI | ∠4 | gra | des | GI : | < 3 | GI | ≥4 | grac | les | 3 | 4 |
| | N % | N % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N % | N % |

Table 11.2.1.7 Itraconazole related Adverse Events. Worst grade per patient

| | _ | P | art A | | | | | | Par | t B | | | | | Par | t A+] | В | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | | | | | | | | | | | | | | | | | | Tota | al |
| | | S1 | (TR | .) | | | S1 (T | R) | | | S2 ( | <u>RT)</u> | | | <u>S1</u> | (TR) | ) | | | |
| | All<br>grades | Cr > 2 | Gr ` | > 1 | A | 11 | Gr | > 2 | Gr | > 1 | A | .11 | Gr | > 2 | Gr | > 1 | A | 11 | Gr 2 | ≥ Gr |
| | grades | OI ≥ 3 | OI 2 | _ + | gra | des | GI | <i>_ 5</i> | GI | < ₹ | gra | des | OI : | _ 3 | OI | <b>∠</b> + | grac | les | 3 | $\geq 4$ |
| | N % | N % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N % | 6 N % |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

<sup>†</sup> Related to both or lurbinectedin or with unknown relationship

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†</sup> Related to both or itraconazole or with unknown relationship

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.2.1.8 Adverse Events regardless of relationship. Worst grade by treatment

| | | | Pa | art A | | |
|--------|------------|------------|------|------------|------|------------|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | Gr≥4 | All grades | Gr≥3 | $Gr \ge 4$ |
| 300/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | | Part B | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | S1 | | | | Sź | 2 | | |
| | T | | R | | R | | | T | |
| SOC/PT | All grades $Gr \ge 3$ | $Gr \ge 4$ All grades | Gr≥3 Gr | $r \ge 4$ All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr≥4 |
| | N(%) N(%) | N(%) N(%) | N(%) N | I(%) N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | Part A- | +B (S1) | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | Т | | | R | | | Total | |
| SOC/PT | All<br>grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 | All grades | $Gr \ge 3$ | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

Table 11.2.1.9 Adverse Events regardless of relationship. Worst grade per patient

| | | | Part 1 | A | | | | | Par | t B | | | | | Par | t A+] | В | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | | | | | | | | | | | | | | | | | | Tota | .1 |
| | | S | 1 (T | R) | | 9 | S1 (7 | ΓR) | | | S2 ( | RT) | | | S1 | (TR | ) | | | |
| | All grades | Gr > 3 | Gr | > 1 | A | .11 | Gr | > 2 | Gr | > 1 | A | .11 | Gr | > 2 | Gr | > 1 | A | 11 | Gr≥ | Gr≥ |
| | grades | OI ≥ 3 | GI | < <del>1</del> | gra | des | GI | <u> </u> | Gi | <b>∠ </b> ₹ | gra | des | OI : | <u> </u> | GI | <b>∠</b> <del>1</del> | grac | des | 3 | 4 |
| | N % | N % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N % | N % |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### Listing 11.2.1.10 AEs grade $\geq 3$

| Study | Sequence | Treatment | Subject | Cycle L | Literal | SOC | PT | Grade | SAE | Start | End | Relationship | Action | Serious Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Part | | Group* | | | term | | | | (Y/N) | date | date | to study | taken | Event |
| | | | | | | | | | | | | medication | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

\* ITZ+LRB / LRB

#### Listing 11.2.1.11 AEs related only to lurbinectedin

| Study Part Sequence Treatment Subject | Cycle | Literal | SOC | PT | Grade | SAE | Start | End | Action | Serious | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group* | | term | | | | (Y/N) | date | date | taken | Event | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

\* ITZ+LRB / LRB

## Listing 11.2.1.12 AEs related only to itraconazole

| Study Part Sequence Treatment Subject | Cycle | Literal | SOC F | PT. | Grade | SAE | Start | End | Action | Serious | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group* | | term | | | | (Y/N) | date | date | taken | Event | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

\* ITZ+LRB / LRB

## 11.2.2 Evolution of Signs and Symptoms during the Treatment

Worst grade of signs and symptoms present at baseline and their evolution during treatment will be shown regardless of relationship.

Table 11.2.2.1 Shift of signs and symptoms during treatment

| 1 able 11.2.2.1 Sillit | of signs and symp | toms u | urmg t | reatifier | 11 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Worst | grade | per pati | ent duri | ng trea | tment | | |
| MedDRA PT | Baseline grade | Gra | de 1 | Grac | le 2 | Grad | de 3 | Gra | de 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | | Part A - | S1 (TR | ) | | | |
| | 1 | | | | | | | | | | |
| | 2 | | | | | | | | | | |
| | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | | | | | | Part B - | S1 (TR | ) | | | |
| | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| ••• | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | | - | | | | Part B - | S2 (RT | ) | | | |
| | 1 | | | | | | | | | | |
| ••• | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test. Test, ITZ+LRB; Reference, LRB alone.

#### 11.3 Serious Adverse Events and Deaths

#### 11.3.1 Serious Adverse Events

This analysis will be carried out on evaluable patients for the safety population.

All serious adverse events tables will be listed by study part and sequence and differentiating by treatment (Test, Reference or both). Additional groups could be done (such as PM01183 alone or in combination) if required, and a sequential number will be added at the end of the table number.

The type of toxicity and worst grade or severity by cycle and by patient will be summarized according to System Organ Class (SOC) and Preferred Term (PT) as per the MedDRA dictionary. Subsequent grouping of similar or clinically related items might be appropriate at the time of the analysis. Tables will be organized by category of events using SOC and PT. Grades could be presented by separate or any other grouping at the time of the analysis.

If the number of SAEs are very low, these tables will not be presented and only listings will be shown.

Table 11.3.1.1 Treatment related<sup>†</sup> (or with unknown relationship) SAEs. Worst grade by treatment

| | | | Pa | art A | | |
|--------|------------|------|------------|------------|------------|------|
| | | T | | | R | |
| SOC/PT | All grades | Gr≥3 | $Gr \ge 4$ | All grades | $Gr \ge 3$ | Gr≥4 |
| 300/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | | | | Par | t B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | S | 1 | | | | | S | 2 | | |
| | | T | | | R | | | R | | | T | |
| SOC/PT | All grades | $Gr \ge 3$ | Gr≥4 | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | Part A- | +B (S1) | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | Т | | | R | | | Total | |
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr ≥ 4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

Table 11.3.1.2 Lurbinectedin related<sup>†</sup> SAEs. Worst grade by treatment

| | | | Pa | ırt A | | |
|---|---|---|---|---|---|---|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | Gr≥4 |
| 500/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | | | | Par | rt B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | S | 1 | | | | | S | 2 | | |
| | | Т | | | R | | | R | | | T | |
| SOC/PT | All<br>grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr ≥ 4 | All<br>grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | Part A- | +B (S1) | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | Т | | | R | | | Total | |
| SOC/PT | All<br>grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr ≥ 4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 11.3.1.3 Itraconazole related<sup>†</sup> SAEs. Worst grade by treatment

| | | | Pa | rt A | | |
|--------|------------|------|------------|------------|------------|------|
| | | T | | | R | |
| SOC/PT | All grades | Gr≥3 | $Gr \ge 4$ | All grades | $Gr \ge 3$ | Gr≥4 |
| 50011 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| ••• | | | | | | |

| | | | | Par | t B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | S1 | | | | | S | 2 | | |
| | T | | R | | | T | | | | |
| SOC/PT | All grades Gr≥3 | $Gr \ge 4$ All grades | $Gr \ge 3$ | Gr≥4 | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr≥4 |
| | N(%) N(%) | N(%) N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | Part A+B (S1) | | | Total | |
|---|---|---|---|---|---|---|
| | T | | R | | Total | |
| SOC/PT | All grades $Gr \ge 3$ | $Gr \ge 4$ All grades | $Gr \ge 3$ $Gr \ge 4$ | All grades | $Gr \ge 3$ | Gr ≥ 4 |

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

| N(%) N(%) N(%) N(%) N | N(%) N(%) | N(%) N(%) |
|-----------------------|-----------|-----------|
|-----------------------|-----------|-----------|

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 11.3.1.4 Treatment related<sup>†</sup> (or with unknown relationship) SAEs. Worst grade per patient

| | <u>.</u> | P | art A | | | | | Par | t B | | | | | Par | t A+ | В | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | | | | | | | | | | | | | | | | | Tota | ĺ |
| | | | (TR | | | | | | | S2 (RT) S1 (TR) | | | | 2) | | | | | |
| | All grades | $Gr \ge 3$ | Gr≥ | <u> 4</u> | All | G | r ≥ 3 | Gr | ≥4 | A | .ll<br>des | Gr | ≥ 3 | Gr | ≥ 4 | All | _ G1 | :≥3 | Gr≥<br>⊿ |
| | N % | | | | | | | | | | | | | | | N S | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Table 11.3.1.5 Lurbinectedin related† SAEs. Worst grade per patient

| | _ | P | art A | | | | | | Part | В | | | | | Par | t A+ | В | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | | | | | | | | | | | | | | | | | | To | otal | |
| | | S1 | (TR | ) | | 5 | S1 (T | R) | | | S2 ( | RT) | | | S1 | (TR | 3) | | | | |
| | All<br>grades | Cr > 2 | Gr > | . 1 | A | .11 | Gr | > 2 | Gr | > 1 | Α | 11 | Gr | > 2 | Gr | > 1 | Α | 11 | Gr > | <sub>2</sub> Gr | `≥ |
| | grades | OI ≥ 3 | Oi ≥ | . + | gra | des | OI | <u> </u> | GI | < <del>'</del> | gra | des | OI : | <u> </u> | OI | <b>∠</b> <del>1</del> | grad | des ' | Ui ≥ | 3 4 | ŀ |
| | N % | N % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N 9 | 6 N | % |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 11.3.1.6 Itraconazole related SAEs. Worst grade per patient

| | | P | art A | | | | | Par | tΒ | | | | | Par | t A+ | -В | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | S1 | (TR) | | | S1 (TI | 5) | | | S2 ( | RT) | | | S1 | (TR | 5) | | Tot | tal |
| | All grades | $Gr \ge 3$ | Gr≥ | 4 gr | All<br>ades | Gr≥ | : 3 | Gr | ≥ 4 | A<br>gra | ll<br>des | Gr | ≥ 3 | Gr | ≥ 4 | Al<br>grad | l<br>les G | r ≥ 3 | 3 Gr≥<br>4 |
| | N % | N % | N % | | % | | % | N | % | N | % | N | % | N | % | | % N | | N % |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†</sup> Related to both or lurbinectedin or with unknown relationship

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†</sup> Related to both or itraconazole or with unknown relationship

T, Test (ITZ+LRB); R, Reference (LRB alone: NA).

Table 11.3.1.7 SAEs regardless of relationship. Worst grade by treatment

| | | | Pa | rt A | | |
|---|---|---|---|---|---|---|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| 300/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | | | Par | t B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | S | 1 | | | | | S | 2 | | |
| | T | T R | | | | | | R | | | |
| SOC/PT | All grades Gr≥3 | Gr≥4 | All<br>grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | Gr≥3 | Gr ≥ 4 |
| | N(%) N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| T R R SOC/PT $\frac{All}{grades}$ $Gr \ge 3$ $Gr \ge 4$ $\frac{All}{grades}$ $Gr \ge 3$ $Gr \ge 4$ All grades $Gr \ge 3$ | Part A+B (S1) Total | Part A+B (S1) | | | |
|---|---|---|---|---|---|
| SOC/PT All $Gr \ge 3$ $Gr \ge 4$ All $Gr \ge 3$ $Gr \ge 4$ All $Gr \ge 3$ $Gr \ge 4$ All $Gr \ge 3$ | R | | Т | | |
| | $Gr \ge 4$ $All grades$ $Gr \ge 3$ $Gr \ge 4$ All grades $Gr \ge 3$ $Gr \ge 4$ | $Gr \ge 4$ g | Gr≥3 | All grades | SOC/PT |
| N(%) | N(%) N(%) N(%) N(%) N(%) N(%) N(%) | N(%) N | N(%) | N(%) | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Table 11.3.1.8 SAEs regardless of relationship. Worst grade per patient

| | _ | P | art A | | | | | | Par | t B | | | | | Par | t A+ | -В | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | | | | | | | | | | | | | | | | | | T | ota | l |
| | | S1 | (TR | ) | | 5 | S1 (T | R) | | | S2 ( | RT) | | | S1 | (TR | (3 | | | | |
| | All<br>grades | Gr > 3 | Gr> | > 4 | A | 11 | Gr | > 3 | Gr | > 1 | A | .11 | Gr | > 3 | Gr | > 4 | A | .11 | Gr > | > 3 ( | Gr≥ |
| | grades | GI <u>~</u> 3 | OI <u>-</u> | - " | gra | des | GI | _ 3 | GI | _ ¬ | gra | des | Gi | _ 3 | Gi | _ ¬ | gra | des | OI <u>-</u> | | 4 |
| | N % | N % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N % |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.3.1.9 All SAEs<sup>†</sup>

| | 9 | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Study | Sequence | Treatment | Subject | SOC | PT Grade | AE Status | AE | AE consequences Start date End date |
| Part | | Group* | | | | | Relationship | |

† SAE narratives will be provided by the pharmacovigilance department

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

S1, Sequence 1; S2, Sequence 2. T, Test (ITZ+LRB); R, Reference (LRB alone).

<sup>\*</sup> ITZ+LRB / LRB

#### 11.3.2 **Deaths**

#### Table 11.3.2.1 Cause of death

| Par | t A | | Pa | rt B | | Part | A+B | _ | |
|---------|-----|------|---------|------|------|------|-----|----|------|
| S1 (TR) | | S1 ( | S1 (TR) | | (RT) | S1 ( | TR) | To | otal |
| N | % | N | % | N | % | N | % | N | % |

Malignant disease

Adverse Event(s)

Other<sup>‡</sup>

Total

Notes: Percentage is based on number of patients who died by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### Listing 11.3.2.2 Deaths

| Study | Sequence Treatment Subj | ect Cycle Death | Cause of | No. of cycles | Time on | Time from first | Time from last |
|---|---|---|---|---|---|---|---|
| Part | Group* | date | death | administered | treatment† | dose (days) | dose (days) |

<sup>\*</sup> ITZ+LRB / LRB

## 11.4 Clinical Laboratory Evaluation

Tables will be listed by study part and sequence, however, additional groups could be done (such as PM01183 alone or in combination) if required, and a sequential number will be added at the end of the table number.

Grades could be presented by separate or any other grouping at the time of the analysis.

## 11.4.1 Hematological Abnormalities

Table 11.4.1.1 Hematological abnormalities: Worst grade by treatment

| | Part A | | | | | |
|---|---|---|---|---|---|---|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | Gr ≥ 4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| Anemia<br>Leukopenia<br>Lymphopenia<br>Neutropenia<br>Thrombocytopenia | | | | | | |

| | Part B | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | S | | | S | 2 | | | | | |
| | T R | | | | | | R | | | Т | |
| SOC/PT | All grades Gr | ≥3 Gr≥4 | All grades | Gr≥3 | Gr ≥ 4 | All grades | Gr≥3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr ≥ 4 |
| | N(%) N( | %) N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Anemia Leukopenia Lymphopenia Neutropenia Thrombocytopenia

| | | | Part A- | -B (S1) | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Т | | | R | | | | |
| SOC/PT | All<br>grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Anemia

Leukopenia

Lymphopenia

Neutropenia

Thrombocytopenia

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

Listing 11.4.1.2 Hematological abnormalities grade  $\geq$  3 by treatment

| Study Part | Sequence | Treatment Group* | Subject | Cycle | Event | Grade |
|------------|----------|------------------|---------|-------|-------|-------|

<sup>\*</sup> ITZ+LRB / LRB

Listing 11.4.1.3 Hematological tests not assessed by treatment

| Study Part | Sequence | Treatment Group* | Subject | Cycle | Lab. test |
|------------|----------|------------------|---------|-------|-----------|

<sup>\*</sup> ITZ+LRB / LRB

Table 11.4.1.4 Hematological abnormalities: Worst grade per patient

| | P | art A | | | Part B | | | Part A+ | В | |
|---|---|---|---|---|---|---|---|---|---|---|
| | C1 | (TD) | | 21 (TD) | c | C2 (DT) | | C1 (TD | ` | Total |
| | | (1K) | | 51 (1K) | | S2 (RT) | | 51 (1K | ) | |
| All<br>grades | $Gr \ge 3$ | $Gr \ge 4$ | All<br>grades | $Gr \ge 3$ | $Gr \ge 4$ | All<br>grades | $Gr \ge 3$ | $Gr \ge 4$ | All<br>grades | $Gr \ge 3 \frac{Gr}{4}$ |
| N % | N % | N % | N % | N % | N % | N % 1 | N % | N % | N % | N % N % |

Anemia

Leukopenia

Lymphopenia

Neutropenia

Thrombocytopenia

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.4.1.5 Hematological abnormalities per patient grade  $\geq 3$ 

| Study Part | Sequence | Treatment<br>Group* | Subject | Cycle | Event | Cycle | Grade |
|---|---|---|---|---|---|---|---|
| ••• | | | | | | | |

<sup>\*</sup> ITZ+LRB / LRB

Listing 11.4.1.6 Hematological tests not assessed per patient

| Study Part | Sequence | Treatment Group* | Subject | Cycle | Lab. test |
|------------|----------|------------------|---------|-------|-----------|

<sup>\*</sup> ITZ+LRB / LRB

#### 11.4.2 Biochemical Abnormalities

Table 11.4.2.1 Biochemical abnormalities: Worst grade per treatment

| | | | 0 1 | | | |
|---|---|---|---|---|---|---|
| | | | Pa | ırt A | | |
| | | T | | | R | |
| | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| ALT increase | | | | | | |
| AST increase | | | | | | |

| | | | | | Par | t B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | S | 51 | | | | | S | 2 | | |
| | Т | | | R | | | R | | | T | |
| All grades | $Gr \ge 3$ | Gr≥4 | All grades | $Gr \ge 3$ | Gr≥4 | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr≥4 |
| N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

ALT increase AST increase

| | | Part A- | +B (S1) | | | | Total | |
|---|---|---|---|---|---|---|---|---|
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | | | Total | | | | | |
| All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr≥4 |
| N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

ALT increase

AST increase

hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia, hypocalcemia.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

Listing 11.4.2.2 Biochemical abnormalities grade ≥ 3 by treatment

| Study Part | Sequence | Treatment Group* | Subject | Event | Grade |
|------------|----------|------------------|---------|-------|-------|

<sup>\*</sup> ITZ+LRB / LRB

Listing 11.4.2.3 Biochemical tests not assessed by treatment

| Study Part | Sequence | Treatment Group* | Subject | Lab. test |
|------------|----------|------------------|---------|-----------|
| ••• | | | | |

<sup>\*</sup> ITZ+LRB / LRB

Notes: Percentage is based on number of patients by study part and sequence, when applicable. \*Creatinine increased, hyperglycemia, hypoglycemia, CPK increased, GGT increased, bilirubin increased,

Table 11.4.2.4 Biochemical abnormalities: Worst grade per patientpatientpatientpatient

| _ | P | art A | | | Part B | | Part A+B | |
|---|---|---|---|---|---|---|---|---|
| | <b>C</b> 1 | (TR) | | 21 (TD) | 52 ( | DT) | S1 (TR) | Total |
| | | | , i | SI (IK) | 52 ( | K1) | | |
| All<br>grades | Gr≥3 | $Gr \ge 4$ | All<br>grades | $Gr \ge 3$ | $Gr \ge 4$ $Gr \ge 4$ $gra$ | $\frac{\text{dl}}{\text{des}} \text{Gr} \ge 3$ | $Gr \ge 4$ $A$ $gra$ | $\frac{.11}{.des} Gr \ge 3 \frac{Gr}{4} \ge$ |
| N % | N % | N % | N % | N % | N % N | % N % | N % N | % N % N % |

ALT increase AST increase ...\*

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.4.2.5 Biochemical abnormalities per patientpatientpatientpatientpatient grade ≥ 3

| Study Part | Sequence | Treatment<br>Group* | Subject | Cycle | Event | Cycle | Grade |
|---|---|---|---|---|---|---|---|

<sup>\*</sup> ITZ+LRB / LRB

Listing 11.4.2.6 Biochemical tests not assessed per patientpatientpatientpatient

| Study Part | Sequence | Treatment Group* | Subject | Cycle | Lab. test |
|------------|----------|------------------|---------|-------|-----------|

<sup>\*</sup> ITZ+LRB / LRB

## 11.4.3 Laboratory Values Over Treatment

Table 11.4.3.1 Shift of hematological abnormalities, worst grade per patient vs. baseline

| Table 11.4.3.1 Si | nift of hematological a | ionormaniies, | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Worst gi | | | | | | | |
| | Baseline grade | Grade 1 | Grade 2 | | Gra | de 3 | Gra | de 4 | Gra | de 5 |
| | | N % | N C | % | N | % | N | % | N | % |
| | | | | P | art A - | S1 (TR | ) | | | |
| Anemia | G0 | - | | | | | | | | |
| | ••• | | | | | | | | | |
| | G4 | | | | | | | | | |
| Leukopenia | G0 | | | | | | | | | |
| | G4 | | | | | | | | | |
| | G0 | | | | | | | | | |
| | ••• | | | | | | | | | |
| | G4 | | | | | | | | | |
| | | | | P | art B - | S1 (TR | ) | | | |
| Anemia | G0 | - | | | | | | | | |
| | ••• | | | | | | | | | |
| | G4 | | | | | | | | | |
| Leukopenia | G0 | | | | | | | | | |
| | G4 | | | | | | | | | |
| ••• | G0 | | | | | | | | | |
| | G4 | | | | | | | | | |
| | | | | P | art B - | S2 (RT | ) | | | |
| Anemia | G0 | | | | | | | | | |
| | G4 | | | | | | | | | |
| Leukopenia | G0 | | | | | | | | | |
| | G4 | | | | | | | | | |
| ••• | G0 | | | | | | | | | |
| | G4 | | | | | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable. Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

If a low number of patients with grade  $\geq 3$  neutropenia or thrombocytopenia, the following table will be omitted and the information will be provided in a listing.

Table 11.4.3.2 Time course for neutrophils and platelets

| | F | Part A | | Part B | | | Part | A+B | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Total |
| | S | 1 (TR) | S1 ( | ΓR) | S2 ( | RT) | S1 ( | (TR) | |
| | N | Median<br>(range) | N | Median (range) | N | Median (range) | N | Median (range) | |
| Neutropenia (Grade≥3) | | | | | | | | | |
| Onset day | | | | | | | | | |
| Nadir day | | | | | | | | | |
| Recovery day | | | | | | | | | |
| Days to recovery | | | | | | | | | |
| Thrombocytopenia (Grade 23) | | | | | | | | | |
| Onset day | | | | | | | | | |
| Nadir day | | | | | | | | | |
| Recovery day | | | | | | | | | |
| Days to recovery | | | | | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.4.3.3 Shift of biochemical abnormalities, worst grade per patient vs baseline

| | | | | Wors | st grade | per pat | ient dur | ing trea | tment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline grade | | de 1 | | de 2 | | ide 3 | | ide 4 | | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | | Part A | · S1 (TR | .) | | | |
| ALT increase | G0 | | | | | | | | | | |
| | <br>G4 | | | | | | | | | | |
| AST increase | G0 | | | | | | | | | | |
| 1151 mereuse | | | | | | | | | | | |
| | G4 | | | | | | | | | | |
| | G0 | | | | | | | | | | |
| | G4 | | | | | Dort D | · S1 (TR | ` | | | |
| A I T : | CO | | | | | Part B | · 51 (1K | .) | | | |
| ALT increase | G0 | | | | | | | | | | |
| | <br>G4 | | | | | | | | | | |
| AST increase | G0 | | | | | | | | | | |
| | G4 | | | | | | | | | | |
| ••• | G0 | | | | | | | | | | |
| | <br>G4 | | | | | | | | | | |
| | | | | | | Part B - | S2 (RT | <u>)</u> | | | |
| ALT increase | G0 | - | | | | | | | | | |
| A CITE : | G4 | | | | | | | | | | |
| AST increase | G0 | | | | | | | | | | |
| | <br>G4 | | | | | | | | | | |
| ••• | G0 | | | | | | | | | | |
| | G4 | | | | | | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

If a low number of patients with grade  $\geq$ 3 ALT or AST increased, the following table will be omitted and the information will be provided in a listing.

Table 11.4.3.4 Time course for AST and ALT

| | Part | A | | P | art B | | Part A+ | В | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 (7 | TR) | S1 ( | TR) | S2 ( | (RT) | S1 (TR | <u>(</u> ) | Тс | otal |
| | N | % | N | % | N | % | N | % | N | % |
| | Part A | * | Pa | rt B | | | :: | Tota | 1 | |
| | | | S1 | (TR) | | S2 (RT) | | | | |
| | N | Med<br>(rang | N | | Median<br>(range) | N | Median (range) | N | | Median range) |
| AST (Grade≥3) | | | | | | | | | | |
| Onset day | | | | | | | | | | |
| Peak day | | | | | | | | | | |
| Recovery day | | | | | | | | | | |
| Days to recovery | | | | | | | | | | |
| ALT (Grade≥3) | | | | | | | | | | |
| Onset day | | | | | | | | | | |
| Peak day | | | | | | | | | | |
| Recovery day | | | | | | | | | | |
| Days to recovery | | | | | | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

### 11.5 Linear Mixed-effects Model

If applicable, to compare the incidence of grade 4 or grade 3/4 between the combination and lurbinectedin alone, a generalized linear mixed-effects model will be fit to the data with treatment (Combination or lurbinectedin alone), period and sequence as fixed effects, and patients nested in sequences as a random effect

Table 11.5.1.1 Safety comparison between combination and lurbinectedin alone<sup>†</sup>

| | Combination | Lurbinectedin alone | p-value <sup>‡</sup> |
|---|---|---|---|
| Any grade 3/4 AE | | | |
| Any grade 4 AE | | | |
| Any grade 3/4 treatment-related AE | | | |
| Any grade 4 treatment-related AE | | | |
| Any abnormality (G3-4) in | | | |
| laboratory value (hema, bio) | | | |
| Any abnormality (G4) in | | | |
| laboratory value (hema, bio) | | | |

<sup>†</sup> A generalized mixed-effects model will be fit for each safety evaluation

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>\*</sup>p-values will be provided for the comparison between treatments (combination vs. Lurbinectedin alone) or including the sequence effect if deemed necessary.

#### 11.6 Physical Findings, ECOG PS, LVEF and ECG

### 11.6.1 Physical Findings and ECOG PS

Listing 11.6.1.1 ECOG Performance status during the study

| C41 | t / C | C1-:4 | | - | PS | | |
|---|---|---|---|---|---|---|---|
| Study | part / Sequence | Subject - | Baseline | Cycle 1 | Cycle 2 | Cycle 3 | EOT |
| Part A | S1 (TR) | | | | | | |
| Part B | S1 (TR) | ••• | | | | | |
| | S2 (RT) | | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.6.1.2 Weight change during the study

| Ctudy n | art / Sequence | Cubicat | Weight (kg) | | % Ch | ange <sup>†</sup> | |
|---|---|---|---|---|---|---|---|
| Study p | art / Sequence | Subject | at baseline | Cycle 1 | Cycle 2 | Cycle 3 | ЕОТ |
| Part A | S1 (TR) | ••• | | | | | |
| Part B | S1 (TR) | ••• | | | | | |
| | S2 (RT) | | | | | | |

<sup>† %</sup> of change with respect to baseline

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.6.1.3 BSA during the study

| Study | art / Saguanaa | Subject — | | | BSA $(m^2)^{\dagger}$ | | |
|---|---|---|---|---|---|---|---|
| Study p | art / Sequence | Subject — | Baseline | Cycle 1 | Cycle 2 | Cycle 3 | EOT |
| Part A | S1 (TR) | | | | | | |
| Part B | S1 (TR) | | | | | | |
| | S2 (RT) | | | | | | |

 $<sup>^{\</sup>dagger}$  Calculated according to DuBois formula: BSA (m<sup>2</sup>) = Weight (kg)<sup>0.425</sup> x Height(cm)<sup>0.725</sup> x 0.007184

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

#### 11.6.2 LVEF and ECG

Listing 11.6.2.1 Patients with abnormal or clinically indicated LVEF during the study

| Study Part Sequence Treatment | Subject | Date | Visit | Abnormal | Specify | Method | LVEF (%) | Lower |
|---|---|---|---|---|---|---|---|---|
| Group* | | | | ity | | | | limit of |
| | | | | | | | | normality |

<sup>\*</sup> ITZ+LRB / LRB

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>\*</sup> ITZ+LRB / LRB

Listing 11.6.2.2 Electrocardiogram: PR interval evolution during the study by study part and sequence

| Study mont / | | PR interval | | | % Change <sup>†</sup> | | |
|---|---|---|---|---|---|---|---|
| Study part / Sequence | Subject | (msec) <sup>‡</sup> at | Сус | ele 1 | Сус | ele 2 | ЕОТ |
| Sequence | | baseline | Pre infusion | Post infusion | Pre infusion | Post infusion | EOI |
| Part A S1 (TR) | | | | | | | |
| Part B S1 (TR) | | | | | | | |
| S2 (RT) | | | | | | | |

<sup>†%</sup> of change with respect to baseline

Listing 11.6.2.3 Electrocardiogram: Heart rate evolution during the study

| C4 1 / | | Heart rate | | | % Change <sup>†</sup> | | |
|---|---|---|---|---|---|---|---|
| Study part /<br>Sequence | Subject | (bpm) <sup>‡</sup> | Сус | ele 1 | Сус | ele 2 | EOT |
| Sequence | | at baseline | Pre infusion | Post infusion | Pre infusion | Post infusion | EOI |
| Part A S1 (TR) | ••• | | | | | | |
| Part B S1 (TR) | | | | | | | |
| S2 (RT) | | | | | | | |

<sup>†%</sup> of change with respect to baseline

Listing 11.6.2.4 Electrocardiogram: QT interval evolution during the study

| C4 1 | , | QT interval | | | % Change <sup>†</sup> | | |
|---|---|---|---|---|---|---|---|
| Study part / Sequence | Subject | (msec) <sup>‡</sup> | Сус | ele 1 | Сус | ele 2 | ЕОТ |
| Sequence | | at baseline | Pre infusion | Post infusion | Pre infusion | Post infusion | |
| Part A S1 (TF | 2) | | | | | | |
| Part B S1 (TF | R) | | | | | | |
| S2 (R7 | T) | | | | | | |

<sup>†%</sup> of change with respect to baseline

<sup>&</sup>lt;sup>‡</sup> Triplicate ECG values obtained at each time point (baseline, Day 1 of Cycle 1 pre-infusion and post-infusion, Day 1 of Cycle 2 pre-infusion and post-infusion and end of treatment) are averaged

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>&</sup>lt;sup>‡</sup> Triplicate ECG values obtained at each time point (baseline, Day 1 of Cycle 1 pre-infusion and post-infusion, Day 1 of Cycle 2 pre-infusion and post-infusion and end of treatment) are averaged

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>&</sup>lt;sup>‡</sup> Triplicate ECG values obtained at each time point (baseline, Day 1 of Cycle 1 pre-infusion and post-infusion, Day 1 of Cycle 2 pre-infusion and post-infusion and end of treatment) are averaged

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.6.2.5 Electrocardiogram: QTc (Bazett's) †† evolution during the study

| | 4/ | | OT- (D#2-)† | | | % Change <sup>†</sup> | | |
|---|---|---|---|---|---|---|---|---|
| Siu | dy part /<br>quence | Subject | QTc (Bazett's) <sup>‡</sup> atbaseline | Сус | ele 1 | Сус | ele 2 | ЕОТ |
| | quence | | at oasciire | Pre infusion | Post infusion | Pre infusion | Post infusion | EOI |
| Part A | S1 (TR) | ••• | | | | | | |
| Part B | S1 (TR) | ••• | | | | | | |
| | S2 (RT) | | | | | | | |

<sup>†%</sup> of change with respect to baseline

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

Listing 11.6.2.6 Patients with abnormal or clinically indicated Electrocardiogram during the study

| StudySequence | Treatment Subject | Cycle Assessm | Visit | ECG #‡ | Result | Specify | PR | Heart | QT | QTc <sup>†</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Part | Group* | ent date | | | | | interval | rate | interval | (Bazett' |
| | | | | | | | (msec) | (bpm) | (msec) | s) |

<sup>†</sup> QTc (Bazett's) = QT interval /  $\sqrt{(60/\text{Heart rate})}$ 

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>&</sup>lt;sup>‡</sup> Triplicate ECG values obtained at each time point (baseline, Day 1 of Cycle 1 pre-infusion and post-infusion, Day 1 of Cycle 2 pre-infusion and post-infusion and end of treatment) are averaged

<sup>††</sup> QTc (Bazett's) = QT interval /  $\sqrt{(60/\text{Heart rate})}$ 

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>\*</sup> ITZ+LRB / LRB

<sup>‡#</sup> of ECGs triplicates: ECG 1-3 (Pre infusion) and ECG 1-3 (Post infusion) identification.

## 11.7 Concomitant Therapies

## 11.7.1 Concomitant Medication during the Study

Table 11.7.1.1 Concomitant medication during treatment (ATC1/ATC2/ATC4/PN)

| Part A | | Par | tB | | | Part A+B | S(S1) | Total |
|--------|-------|-------|-------|-------|-------|----------|-------|-------|
| T | R | T | R | T | R | T | R | |
| N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |
| ATC1 | | | | | | | | |
| ATC 2 | | | | | | | | |
| ATC4 | | | | | | | | |
| PN | | | | | | | | |
| 4TC1 | | | | | | | | |
| ATC 2 | | | | | | | | |
| ATC4 | | | | | | | | |
| PN | | | | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.7.1.2 Concomitant medication during treatment by ATC

| Par | t A | | Pai | rt B | | Part A- | +B (S1) | |
|---|---|---|---|---|---|---|---|---|
| T | R | T | R | T | R | T | R | Total |
| N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |
| No. of system | ıs (ATC1 lev | rel) | | | | | | |
| 0 | | | | | | | | |
| 1 | | | | | | | | |
| 2<br>≥ 3 | | | | | | | | |
| ≥ 3<br>Median (rang | TO) | | | | | | | |
| No. of indicar | | level) | - | | | | | |
| $\theta$ | nons (ATC2 | ievei) | | | | | | |
| i<br>1 | | | | | | | | |
| 2 | | | | | | | | |
| ≥ <i>3</i> | | | | | | | | |
| Median (rang | ge) | | | | | | | |
| No. of agent | | C4 level) | - | | | | | |
| 0 | ` | ŕ | | | | | | |
| 1 | | | | | | | | |
| 2 | | | | | | | | |
| ≥ <i>3</i> | | | | | | | | |
| Median (rang | | | - | | | | | |
| No. of agents | (PN level) | | | | | | | |
| 0 | | | | | | | | |
| 1 | | | | | | | | |
| 2 | | | | | | | | |
| ≥3<br>Madian (nana | ra) | | | | | | | |
| Median (rang | (e) | | | | | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.7.1.3 Summary of concomitant medication during treatment by ATC

| Par | rt A | | Par | rt B | | Part A- | +B (S1) | |
|---|---|---|---|---|---|---|---|---|
| T | R | T | R | Т | R | T | R | Total |
| N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |
| No. of systen | ns (ATC1 lev | rel) | | | | | | |
| N | • | | | | | | | |
| Median (ran | ge) | | | | | | | |
| No. of indica | tions (ATC2 | level) | | | | | | |
| N | ` | , | | | | | | |
| Median (ran | ge) | | | | | | | |
| No. of agent | families (AT | C4 level) | : | | | | | |
| N | | , | | | | | | |
| Median (ran | ge) | | | | | | | |
| No. of agents | <del>-</del> | | | | | | | |
| N | , | | | | | | | |
| Median (ran | ge) | | | | | | | |
| | 4 14 | C 1 | D / D | • | 1 1 1 | | | |

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

## 11.7.2 Further Antitumor Therapies

Listing 11.7.2.1 First Antitumor Therapy

| Study Part | Sequence | Subject | End of treatment | First Antitumor<br>Therapy | Start date |
|---|---|---|---|---|---|

<sup>\*</sup> ITZ+LRB / LRB

# 12 APPENDIX III: EFFICACY EVALUATION

Not applicable.

# 13 APPENDIX IV: DB Listings

| Listing 13.1 Scr | eening (I) | | | | | |
|---|---|---|---|---|---|---|
| | | l PGt sub- Pla | • | | 3 EC4 PCR P | |
| Sequence | consent | study initi | ation type | prior lines | date re | sult |
| Listing 13.2 Scr | eening (II) | | | | | |
| Part / Sequence | | Subject | Screening failure | Criterion | not met | Details |
| Turr soquen | | | zereeming iumure | | | |
| Listing 13.3 Spo | nsor Approv | val Form | | | | |
| Part / Sequen | | oject Approv | val Comments S | Study Part Lurl | binectedin in Lur | binectedin alone |
| _ | | | | | ombination | (mg/m2) |
| | | | | | (mg/m2) | |
| T 12.4 D | 1 | 1 . 11 | | | | |
| Listing 13.4 Ran | | | J., 4. 1 | -4 | Danaminatian | D-4-/T: |
| Part / Sequence | Subje | | , | atment ]<br>uence | Description | Date/Time |
| | | Tanc | ionnized Seq | uchec | | |
| Listing 13.5 Stud | dy registratio | on | | | | |
| Part / | Subject | Registration | Randomization | Sequence | Description | Screening |
| Sequence | Subject | registration | Tundonnzunon | Sequence | Bescription | failure date |
| | | | * | | | • |
| Listing 13.6 Dat | e of visit | | | | | |
| Part / Sequence | Treatment ( | Group* Su | ibject C | ycle | Visit | Date |
| Part / Sequence * ITZ+LRB / LRB | | Group* Su | ibject C | ycle | Visit | Date |
| | | Group* Su | ibject C | ycle | Visit | Date |
| | 3 | • | ıbject C | ycle | Visit | Date |
| * ITZ+LRB / LRE | 3 | • | Cycle | ycle Visit | Visit | Date Clinically |
| * ITZ+LRB / LRE<br>Listing 13.7 Dat<br>Part / Sequence | e of unsched<br>Treatment<br>Group* | luled visit | | | | Clinically |
| * ITZ+LRB / LRE<br>Listing 13.7 Dat | e of unsched<br>Treatment<br>Group* | luled visit | | | | Clinically |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE | e of unsched<br>Treatment<br>Group* | luled visit | | | | Clinically |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der | e of unsched<br>Treatment<br>Group* | luled visit<br>Subject | Cycle | | | Clinically |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE | e of unsched<br>Treatment<br>Group* | luled visit | Cycle | | | Clinically indicated repeat |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der | e of unsched<br>Treatment<br>Group* | luled visit<br>Subject | Cycle | Visit | Date | Clinically<br>indicated repeat |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der | e of unsched<br>Treatment<br>Group* | luled visit<br>Subject | Cycle | Visit | Date | Clinically indicated repeat |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence | e of unsched<br>Treatment<br>Group*<br>3<br>nographics<br>Subject | luled visit Subject Date of birt | Cycle h Age (years) | Visit | Date | Clinically indicated repeat |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi | e of unsched Treatment Group* nographics Subject | luled visit Subject Date of birt | Cycle h Age (years) | Visit<br>Sex | Date<br>Race | Clinically indicated repeat Other Race, specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence | e of unsched<br>Treatment<br>Group*<br>3<br>nographics<br>Subject | Date of birt | Cycle h Age (years) equate contraception bearing No, 1 | Visit Sex On Reason | Date Race | Clinically indicated repeat |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi | e of unsched Treatment Group* nographics Subject | Date of birt | Cycle h Age (years) | Visit Sex On Reason | Date<br>Race | Clinically indicated repeat Other Race, specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi | e of unsched Treatment Group* nographics Subject | Date of birt | Cycle h Age (years) equate contraception bearing No, 1 | Visit Sex On Reason | Date Race | Clinically indicated repeat Other Race, specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi Part / Sequence | e of unsched<br>Treatment<br>Group*<br>Inographics<br>Subject | Date of birt | Cycle h Age (years) equate contraception bearing No, 1 | Visit Sex On Reason | Date Race | Clinically indicated repeat Other Race, specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi Part / Sequence Listing 13.10 Pr | e of unsched Treatment Group* nographics Subject Idbearing po Subje | luled visit Subject Date of birt otential and addet Child | Cycle h Age (years) equate contraception bearing No, I ential? | Visit Sex on Reason | Pate Race Adequate ontraception? | Clinically indicated repeat Other Race, specify Specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi Part / Sequence Listing 13.10 Property | e of unsched<br>Treatment<br>Group*<br>Inographics<br>Subject | Date of birt | Cycle h Age (years) equate contraception bearing No, I ential? | Visit Sex On Reason | Date Race | Clinically indicated repeat Other Race, specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi Part / Sequence Listing 13.10 Pr | e of unsched Treatment Group* nographics Subject Idbearing po Subje | luled visit Subject Date of birt otential and addet Child | Cycle h Age (years) equate contraception bearing No, I ential? | Visit Sex on Reason | Pate Race Adequate ontraception? | Clinically indicated repeat Other Race, specify Specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi Part / Sequence Listing 13.10 Property | e of unsched Treatment Group* nographics Subject Idbearing po Subje | luled visit Subject Date of birt otential and addet Child | Cycle h Age (years) equate contraception bearing No, I ential? | Visit Sex on Reason | Pate Race Adequate ontraception? | Clinically indicated repeat Other Race, specify Specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi Part / Sequence Listing 13.10 Property / Sequence | e of unsched Treatment Group* nographics Subject Idbearing po Subject egnancy test Subject | Date of birt otential and added Ct Not applicable | Cycle h Age (years) equate contraception bearing No, I ential? | Visit Sex on Reason | Pate Race Adequate ontraception? | Clinically indicated repeat Other Race, specify Specify |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi Part / Sequence Listing 13.10 Property of the part / Sequence Listing 13.11 Property of the part / Sequence | e of unsched Treatment Group* nographics Subject Idbearing po Subject Subject Subject Subject | Date of birt otential and addet Child pot Not applicable | Cycle h Age (years) equate contraception ibearing No, 1 ential? e? Reason | Visit Sex On Reason Co Not done? | Date Race Adequate ontraception? Sample date | Clinically indicated repeat Other Race, specify Specify Result |
| * ITZ+LRB / LRE Listing 13.7 Dat Part / Sequence * ITZ+LRB / LRE Listing 13.8 Der Part / Sequence Listing 13.9 Chi Part / Sequence Listing 13.10 Property Sequence Listing 13.11 Property Sequence | e of unsched Treatment Group* nographics Subject Idbearing po Subje egnancy test Subject | Date of birt otential and added Ct Not applicable | Cycle h Age (years) equate contraception bearing No, I ential? | Visit Sex On Reason Co Not done? | Date Race Adequate ontraception? Sample date | Clinically indicated repeat Other Race, specify Specify Result |

| Listing 13.12 Canc | er history |
|--------------------|------------|
|--------------------|------------|

| Listing 13.12 | 2 Cancer hist | ory | | E' 4 1' | | | 1' |
|---|---|---|---|---|---|---|---|
| Part / | C1-:4 | Date of | Т | First dia | | Current of | |
| Sequence | Subject | diagnosis | Tumor type | Stage | Date of advanced disease | metastatic disease | |
| * ITZ+LRB / | LRB | | | | <u> </u> | | · |
| Listing 13.13 | 3 Prior surger | <b>:</b> V | | | | | |
| Part / Seq | | Subject | | None? | Site and | procedures | Date |
| Listing 13.1 | 4 Prior radiot | herapy | | | | | |
| Part /<br>Sequence | Subject | None? | Site | Total dos<br>(Gy) | e Date o | of first dose D | ate of last dose |
| Sequence | | | , | (Gy) | | | |
| I : .: 12.1. | 7 D : | 1. | 1.4 | | | | |
| Listing 13.1;<br>Part / | 5 Prior antica<br>Subject | | | n Agent A | gent Agent | Setting Start Stop | Best PD N |
| Sequence | Buoject | , 1 | one: Regime | | oded Class | | response date I |
| | | | | | · | | |
| Listing 13.10 | 6 Prophylacti | c medicatio | n | | | | |
| | | | | Route Dail | y Units Sta | art Stop Time Ta | ken per Speci |
| Sequence | VC2 ATC2 AT | PC/4 | | dose | e da | te date pr | rotocol |
| * ITZ+LRB / | C2, ATC3, AT<br>LRB | 104 | | | | | |
| Listing 13.1 | 7 Lurbinected | lin administ | ration | | | | |
| | tment Subject | Cycle Visit | | | | Total Total | Total BSA |
| Sequence Gro | oup* | | | time time | | ntended dose ose (mg) given | volume calcula<br>for do |
| * ITZ+LRB / | LRB | · | | | (mg/mz) a | ose (mg) given | 101 40 |
| Listing 13 1 | 8 Lurbinected | lin treatmen | t modificatio | n | | | |
| | eatment Subje | | | | fication 1 | Reason Adver | se Other, |
| Sequence G | | | modific | ation | | Even | t specify |
| Listing 13.19 | 9 Lurbinected | lin re-admir | istration | | | | |
| | atment Subject | t Cycle | Visit Dat | te Not do | ne? Route | | rt time End tin |
| Sequence Gro<br>* ITZ+LRB / | | | | | | given | |
| | 0 Itraconazol | | | | | | |
| Part / Trea<br>Sequence t Gr | atmen Subject | Cycle V <sub>1S1</sub> | t Day Date | | | Faken R<br>secordingly? | eason Contac |
| * ITZ+LRB / | | b | | | poures | io o o rumgij i | |
| T :-4: 12 2: | 1 14 | 4::-4 | 4: D1 4 - D | o | | | |
| | 1 Itraconazolatmen Subject | | | | o. of | Γaken R | eason Contac |
| Sequence t Gr | - | | | | | accordingly? | |
| * ITZ+LRB / | LRB | | | | | | |
| Listing 13.22 | 2 Hematologi | ical laborato | ry values | | | | |
| | atmentSubject | CRF Calc. I<br>Visit cycle | - | | | utrophils Lymphoc<br>10*9/L) (x10*9/ | • |
| Sequence Gro (†)Hematocrit | oup*<br>, RBC and mo | | (g/dl) | (X | 10.9/L) (X | 10.3/L) (X10.49/ | L) (x10*9/I |
| * ITZ+LRB / | | J | | | | | |

| Part /<br>Sequence | Treatment<br>ce Group* | Subject | Cycle | Vi | sit Calcula<br>cycle | | Repeat | INR (ratio) |
|---|---|---|---|---|---|---|---|---|
| * ITZ+LF | RB / LRB | | | | | | | |
| | 3.24 Biocher | | _ <u></u> | | | | | |
| Part / T<br>Sequen<br>ce | Freatment Subj<br>Group* | | ilc. Date | n T | otal Bilirubin<br>(mg/dl) | Direct<br>Bilirubin<br>(mg/dl) | AST ALT (IU/L) (IU/L | |
| Acid Gly | ine, CrCl, Glucoprotein, Inter<br>RB / LRB | | PK-MB fr | action, G | GT, Total Proto | | n, CRP, Na, K | , Mg, Ca, Alpha-1- |
| | 3.25 Perform | | . , | G 1 | N 1 | T7' '. | D / | FCOC |
| Part A<br>Sequer | | | ject | Cycle | Not done | Visit | Date | ECOG |
| 112.121 | XD / LKD | | | | | | | |
| | 3.26 Physica | | | 71 1. 5 | | 11. 501 | DG. | <del></del> |
| | Treatment Su<br>Group* | bject Cycle | Not V<br>done | /isit Dat | te Weight Hei | ight BSA<br>method | | Any Findings malities? |
| (istina 1 | 2 27 Wital air | | | | | | | |
| Part / | 3.27 Vital sig | | cle Not | done | Visit Date | Heart rat | e Systolic Γ | Diastolic Temperat |
| Sequence | | ineget eg | 1100 | 40114 | . 1510 | | | |
| | e Group* | | | | | (bpm) | (шшпо) (1 | mmHG) ure (°C) |
| | RB / LRB | | <u> </u> | | | (opm) | (DHIIII) | mmHG) ure (*C) |
| * ITZ+LF | RB / LRB | cardiogram | | | | (opm) | (mino) (i | mmHG) ure (°C) |
| * ITZ+LF<br>Listing 1 | RB / LRB 3.28 Electroceatment Subjection | | Date # | Pre/P No | ot Result Spec | | Heart QT<br>rate interval | Bazett's Not done corrected within QT protocol, |
| * ITZ+LF<br>Listing 1<br>Part / Tr<br>Seque C<br>nce | RB / LRB 3.28 Electroceatment Subjectroup* | | Date # | | | ify PR interval | Heart QT<br>rate interval | Bazett's Not done corrected within |
| * ITZ+LF<br>Listing 1<br>Part / Tr<br>Seque C<br>nce | RB / LRB 3.28 Electroceatment Subjection | | Date # | | | ify PR interval | Heart QT<br>rate interval | Bazett's Not done corrected within QT protocol, |
| * ITZ+LF<br>Listing 1<br>Part / Tr<br>Seque C<br>nce | RB / LRB 3.28 Electroceatment Subjectroup* | etCycle Visit | iagnostic | ost dor | ne | ify PR interval | Heart QT<br>rate interval | Bazett's Not done corrected within QT protocol, |
| Listing 1 Part / Tr Seque Conce ITZ+LF Listing 1 Part / | RB / LRB 3.28 Electroc eatment Subjection Froup* RB / LRB 3.29 Concon Treatmen | etCycle Visit | iagnostic | ost dor | res | ify PR interval (msec) ( | Heart QT<br>rate interval | Bazett's Not done corrected within QT protocol, specify |
| Listing 1 Part / Tr Seque C nce * ITZ+LF Listing 1 Part / Sequen | RB / LRB 3.28 Electroceatment Subjections RB / LRB 3.29 Concon Treatmen Group* | etCycle Visit | iagnostic | ost dor | res | ify PR interval (msec) ( | Heart QT<br>rate interval<br>bpm) (msec) | Bazett's Not done corrected within QT protocol, specify |
| Listing 1 Part / Tr Seque C nce * ITZ+LF Listing 1 Part / Sequence * ITZ+LF | RB / LRB 3.28 Electroceatment Subjections RB / LRB 3.29 Concon Treatment Group* RB / LRB | etCycle Visit | iagnostic | ost dor | res | ify PR interval (msec) ( | Heart QT<br>rate interval<br>bpm) (msec) | Bazett's Not done corrected within QT protocol, specify |
| Listing 1 Part / Tr Seque C nce ITZ+LF Listing 1 Part / Sequence ITZ+LF | RB / LRB 3.28 Electroceatment Subjections RB / LRB 3.29 Concom Treatment Ce Group* RB / LRB 3.30 LVEF | nitant non-d | iagnostic<br>Cycl | procedu<br>e Pro | res<br>ocedure D | ify PR interval (msec) ( | Heart QT rate interval bpm) (msec) | Bazett's Not done corrected within QT protocol, specify MH Comments |
| Listing 1 Part / Tr Seque Conce * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Part / | RB / LRB 3.28 Electroceatment Subjections RB / LRB 3.29 Concon Treatment Group* RB / LRB | nitant non-d | iagnostic | procedure Pro | res | ify PR interval (msec) ( | Heart QT rate interval bpm) (msec) | Bazett's Not done corrected within QT protocol, specify |
| Listing 1 Part / Tr Seque Conce ITZ+LF Listing 1 Part / Sequence ITZ+LF Listing 1 Part / Sequence | RB / LRB 3.28 Electroceatment Subjections* RB / LRB 3.29 Concom Treatment Ce Group* RB / LRB 3.30 LVEF Treatment Subjections | nitant non-d | iagnostic<br>Cycl<br>Reason<br>clinically | procedure Pro | res<br>ocedure D | ify PR interval (msec) ( | Heart QT rate interval bpm) (msec) cation AE/ | Bazett's Not done corrected within QT protocol, specify MH Comments Result Abnorm al |
| Listing 1 Part / Tr Seque Conce ITZ+LF Listing 1 Part / Sequence ITZ+LF Listing 1 Part / Sequence ITZ+LF | RB / LRB 3.28 Electroceatment Subjects RB / LRB 3.29 Concon Treatment Group* RB / LRB 3.30 LVEF Treatment Subjects Group* | nitant non-d<br>t Subject | iagnostic<br>Cycl<br>Reason<br>clinically<br>indicated | procedure Pro | res<br>ocedure D | ify PR interval (msec) ( | Heart QT rate interval bpm) (msec) cation AE/ | Bazett's Not done corrected within QT protocol, specify MH Comments Result Abnorm al |
| Listing 1 Part / Tr Seque Conce ITZ+LF Listing 1 Part / Sequence ITZ+LF Listing 1 Part / Sequence ITZ+LF | RB / LRB 3.28 Electroce eatment Subject Group* RB / LRB 3.29 Concom Treatment Group* RB / LRB 3.30 LVEF Treatment Subject Group* RB / LRB 3.31 Signs and Signs are suppressed in the subject Group* | nitant non-d t Subject | Reason clinically indicated | procedure Pro | res ocedure D | ify PR interval (msec) ( | Heart QT rate interval bpm) (msec) cation AE/ | Bazett's Not done corrected within QT protocol, specify MH Comments Result Abnorm al specify |
| Listing 1 Part / Tr Seque Conce * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence | RB / LRB 3.28 Electroceatment Subjections RB / LRB 3.29 Concom Treatment Ce Group* RB / LRB 3.30 LVEF Treatment Subjections Group* RB / LRB 3.31 Signs at Treatment Subjections Group* | nitant non-d t Subject | Reason clinically indicated | procedure Pro | res ocedure D | ify PR interval (msec) ( | Heart QT rate interval bpm) (msec) cation AE/ | Bazett's Not done corrected within QT protocol, specify MH Comments Result Abnorm al |
| Listing 1 Part / Tr Seque Conce * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 | RB / LRB 3.28 Electroce eatment Subject Group* RB / LRB 3.29 Concom Treatment ce Group* RB / LRB 3.30 LVEF Treatment Subject Group* RB / LRB 3.31 Signs and Treatment Subject Group* | nitant non-d t Subject | Reason clinically indicated | procedure Pro | res ocedure D Visit Date Ong. End Ong | ify PR interval (msec) ( | Heart QT rate interval bpm) (msec) cation AE/ | Bazett's Not done corrected within QT protocol, specify MH Comments Result Abnorm al specify |
| * ITZ+LF Listing 1 Part / Tr Seque Conce * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence * ITZ+LF Listing 1 Part / Sequence | RB / LRB 3.28 Electroceatment Subjections RB / LRB 3.29 Concom Treatment CE Group* RB / LRB 3.30 LVEF Treatment Subjections Group* RB / LRB 3.31 Signs and Treatment Subjections Group* MedDRA PT | nitant non-d t Subject bject Cycle ad symptom | Reason clinically indicated | procedure Pro | res ocedure D Visit Date Ong. End Ong | ify PR interval (msec) ( | Heart QT rate interval bpm) (msec) cation AE/ | Bazett's Not done corrected within QT protocol, specify MH Comments Result Abnorm al specify |

| Listing 13.33 SAE summary | | | | | | |
|---|---|---|---|---|---|---|
| Part / Treatme Subject Case id. | AE† Outc | ome Start Deat | | | | o Discharge‡ |
| Sequen nt<br>ce Group* | | date | threatenin<br>g | hospitalizati | n date | date |
| (†)SOC, MedDRA PT<br>(‡)Persistent/significant disability/in<br>agent transmitted, narrative, nullific<br>* ITZ+LRB / LRB | | nital anomaly, o | other medica | on<br>lly important | serious e | event, infectious |
| Listing 13.34 Concomitant med | | | | | | |
| Part / Treatment Subject Cycle<br>Sequen Group* | Medication <sup>†</sup> | Route Dose (units) | | Start End On<br>date date | going Inc | lication AE/MH |
| (†)ATC1, ATC4<br>* ITZ+LRB / LRB | | | | | | |
| Listing 13.35 Diagnostic proced | | | | | | |
| Part / Treatment Subject Sequence Group* * ITZ+LRB / LRB | ct Cycle | Test | Date | Result | Units | Comments |
| Listing 13.35.1 Pharmacokinetic | es | | | | | |
| Part / Treatme Subject Cycle<br>Sequen nt | | Samp. Date vindow | | otal Unboun<br>one) d (done) | ites | Itracona Comme<br>zole nts |
| ce Group* * ITZ+LRB / LRB | · | · | · | <u> </u> | (done) | (done) |
| Listing 13.36 Alpha-1-acid glyc | conrotein and Ir | nterleukin 6 | | | | |
| Part / Sequence Treatment | Subject | Visit | Sample tal | ken Da | ate | Comments |
| Group* * ITZ+LRB / LRB | | | - | | | |
| Listing 13.37 Pharmacogenetics | s (Polymorphis | ms) | | | | |
| Part / Sequence Subject | Cycle | | Date | Not done | ? | Comments |
| Listing 13.38 End of treatment Part / Sequence | Subject | Prim | ary Reason I | End of | Sr | pecify |
| - art sequence | Subject | | Treatment | | 51 | |
| Listing 13.39 Follow up - Furth | | | | | C. | . 1 . |
| Part / Sequence | Subject | An | titumor The<br>description | | Sta | rt date |
| Listing 13.40 Off study | | | | | | |
| Part / Sequence Max. Cycle received | Subjec | et ] | Date | Primary rea | son | Specify |
| Listing 13.41 Death report form | | . D 41.1 | | | | A 4 9 |
| Part / Sequence Max. Cycle receiv | ved Subjec | t Death da | ate Cau | ise Sp | pecify | Autopsy? |
| Listing 13.42 Investigator comm | nents | | | | | |
| Part / Sequence Treatment Group* | Subject | Page name | Instance | e Var | iable | Comments |
| * ITZ+LRB / LRB | · | | | | | |
### 14 APPENDIX V: BIMO Listings

The following listings will be provided following the recommended standardized formats according to the draft Guidance for Industry Standardized Format for Electronic Submission of NDA and BLA Content for the Planning of Bioresearch Monitoring (BIMO) Inspections for CDER Submissions (February 2018) and the associated Bioresearch Monitoring Technical Conformance Guide Containing Technical Specifications.

https://www.fda.gov/downloads/Drugs/DevelopmentApprovalProcess/FormsSubmissionRequirements/UCM332466.pdf

https://www.fda.gov/downloads/Drugs/DevelopmentApprovalProcess/FormsSubmissionRequirements/UCM332468.pdf

| Table 14.1 Site lev | el summary | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site | | Patie<br>Scree | | | | atients End<br>Treatmen | P | Patients Off Study | |
| I :-4: 142 C | 4 . 4 1 4 . | - 1:4- | | | | | | | |
| Listing 14.2 Conse | | s by site | | | | | | | D . C |
| Part / Site Sequenc | Treatment<br>e Group* | Subject | Infor<br>Conse | | Screening failure? | Date<br>Screen<br>failu | ning T | reated | Date of<br>First<br>treatment |
| * ITZ+LRB / LRB | | | | | | | | | |
| Listing 14.3 Seque | ence assignme | ent by site | | | | | | | |
| Site | Subject | | Stud | dy Part | | | tment<br>ience | First | Intended<br>dose |
| Listing 14.4 Disco | End of | treatment | ] | | reatment, | Off-stu | • | study | Off-study |
| | Re | eason | | spo | ecify | date | : Re | ason | Specify |
| Listing 14.5 Study | population b | y site | | | | | | | |
| Site Subject | Enrolled p | opulation | PK po | pulation | n Reas | on Sa | fety popula | ation | Reason |
| Listing 14.6 Inclus | | | | | | | | | |
| Site Si | ıbject | Eligibility 1 | equirem | ents? | Cr | iterion ider | ntifier I/E | | I/E details |
| Listing 14.7 Adver | | | | | | | | | |
| Site Subject | Adverse<br>Event | ICI-<br>CTC SAE<br>rade | Onset<br>date | End<br>date | Relationship<br>Specify | Action taken | Seriousn<br>Criteri | | Outcome |
| Listing 14.8 Death | s by site | | | | | | | | |
| Site | Subject | | Date | | Reaso | | Fime from<br>first dose<br>(days) | | ne from last<br>ose (days) |

| †ATC1, ATC4 Listing 14.11 Individual Laboratory Measurements by site Site Subject Cycle Examinatio n date Laboratory Hematocri t RBC (x10*9/L) ls (x10*9/L) (x10*9/L) ls (x10*9/L) (x10*9/L) ls (x10*9 | | | Site | | | | Subject | | Deviation t | ype | | De | evia |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| type Medication Reason interval date date interval type Medication Reason interval date date interval type Medication Reason interval date date interval type interval date date date interval date date date date interval date | Listin | g 14.10 Cc | oncomita | nt med | ication | | | | | | | | |
| Listing 14.11 Individual Laboratory Measurements by site Site Subject Cycle Examinatio n date Laboratory Hematocri t RBC WBC (x10*9/L) Is (x10*9/L) (x10*9/ | Site | Subject M | | Medic | ation F | Reason | † Rou | | | | | Indication | A |
| Site Subject Cycle Examinatio n date Laboratory Hematocri t RBC WBC (x10*9/L) ls (x10*) *Lymphocytes, Monocytes, Platelets, INR, Creatinine, CrCl, Glucose, CPK, CPK-MB fraction, GGT Albumin, CRP, Na, K, Mg, Ca, Alpha-1-Acid Glycoprotein, Interleukin 6. *Listings 14.12 Electrocardiogram by Site* Site Subject Visit Date ECG# Not Result Specify PR Heart QT interval rate interval compact (msec) (bpm) (msec) Compact (msec) (bpm) (msec) Compact (msec) (bpm) ( | †ATC1 | , ATC4 | | | | | | | | | | | |
| Site Subject Cycle Examination date Laboratory t RBC (x10*9/L) ls (x10*9/L) (x10*9/L) ls (x10*9/ | Listin | g 14.11 Inc | dividual | Labora | tory Me | easuren | nents by s | ite | | | | | |
| Albumin, CRP, Na, K, Mg, Ca, Alpha-1-Acid Glycoprotein, Interleukin 6. Listings 14.12 Electrocardiogram by Site Site Subject Visit Date ECG# Not Result Specify PR Heart QT interval rate interval compact (msec) (bpm) (msec) Listings 14.13 LVEF by Site Site Subject Visit Date Not Done Method LVEF (%) Range Abnormality Site Subject Visit Date Not Done Method LVEF (%) Range Range Not Done Method LVEF (%) Range R | Site | Subject | Cycle | | inatio I | aborato | orv | tocri | RBC (x | | τ.) | eutrophi<br>ls<br>10*9/L) | |
| Listings 14.12 Electrocardiogram by Site Site Subject Visit Date ECG# Not Result Specify PR Heart QT Einterval rate interval compact (msec) (bpm) (msec) Listings 14.13 LVEF by Site Site Subject Visit Date Not Done Method LVEF (%) Range Abnormality Site | | • | | | | | | | | MB frac | ction, C | GT, Total | Pr |
| Site Subject Visit Date ECG# Not Result Specify PR Heart QT Interval rate interval compact (msec) (bpm) (msec) Compact | Aloum | iin, CKP, N | a, K, Mg, | Ca, Alp | na-1-Ac | ia Glyc | oprotein, i | nterieukin | 0. | | | | |
| Listings 14.13 LVEF by Site Site Subject Visit Date Not Done Method LVEF (%) Range Abnormality S | Listin | gs 14.12 E | lectrocai | diograi | n by Si | te | | | | | | | |
| Site Subject Visit Date Not Done Method LVEF (%) Range Abnormality S | | Subject | Visit | Date | ECG# | Not | Result | Specify | PR H | | - | Bazett's | ľ |
| Site Subject Visit Date Not Done Method LVEF (%) Range Abnormality S | Site | Subject | | | | done | | | | | | l correcte<br>QT | ŗ |
| Site Subject Visit Date Not Done Method LVEF (%) Range Abnormality S | Site | Subject | | | · | done | | | | | | | d v |
| | | | VEF by | Site | - | done | | | | | | | ŗ |
| Lower<br>Limit | Listin | gs 14.13 L | | | Not Do | | Method | LVEF ( | (msec) (b | opm) ( | (msec) | QT | I s |

Repeat

# 15 APPENDIX VI: ICH Listings

In accordance with the ICH E-3 guideline, patient listings specified as section 16.2 will be prepared.

| 1 1 |
|---|
| Listing 16.2.1 Discontinued Patients |
| Part / Treatment First Last Reason for |
| Sequence Group* Subject Institution Treated Cycles received receiv |
| date date treatment |
| * ITZ+LRB / LRB |
| Listing 16.2.2 Protocol Deviations |
| Subject Deviation type Description |
| Listing 16.2.3 Patients excluded from the efficacy analysis |
| Not applicable |
| Listing 16.2.4 Demographic data |
| Subject Tumor Stage <sup>†</sup> Age Gender Race ECOG Weight Height BSA Prior Prior Prior |
| type (kg) (cm) (m²) radiotnerapy surgery agents |
| †At diagnosis |
| Listing 16.2.5 Compliance and/or drug concentration data |
| Lurbinectedin Itraconazole |
| Subject First Start Start Total dose (First (Second dose (First (Second (mg/m²/ mg/m²/ intensity dose (mg/m²/ inte |
| (mg/m2) cycle) cycle) wk) (%) |
| †Delays/reductions will be nested for each patient (cycle and reason of delay/reduction), e.g. C2 hematological toxicity |
| toxicity |
| Listing 16.2.6 Individual efficacy response data |
| Not applicable |
| Listing 16.2.7 Adverse Event listing (each patient) |
| Subject Adverse Event SOC PT Grade SAE Onset End date date Relationship Action Seriousness Outcome |
| Listing 16.2.8 Individual Laboratory Measurements by Patient |
| Hematocrit RBC $\frac{\text{WBC}}{(\text{x}10*9/\text{L})} \frac{\text{Neutrophils}}{(\text{x}10*9/\text{L})} \cdots^{\dagger}$ |
| Subject Cycle Examination date Laboratory Std. value Std. value Std. value Std. value Std. value Std. value |
| *Lymphocytes, Monocytes, Platelets, INR, Creatinine, CrCl, Glucose, CPK, CPK-MB fraction, GGT, Total Proteins, |
| Albumin, CRP, Na, K, Mg, Ca, Alpha-1-Acid Glycoprotein, Interleukin 6. |

#### 15.1 History of Changes

Clarifications and modifications have been added to the SAP v2.0 on date 25 May 2022.

A summary of such changes are include below:

- 1. On Appendix I (Patients Disposition) columns and footnotes to the tables and listings have been included in order to clarify. See below (\*).
- 2. On Appendix II (Safety Analysis) some tables headers have been clarified and updated. Also new footnotes have been included. See below (\*\*).
- 3. On Appendix IV (DB Listings) columns Treatment Group and Cycle have been included, where applicable. See below (\*\*\*).

Changes are presented in the following pages. Inclusions are highlighted in *Italic bold* and text removed has been <del>crossed out</del>. Minor corrections will not be described below.

### (\*) Appendix I (Patients Disposition)

#### All Sections

On tables 10.1.1.1, 10.1.1.3, 10.1.2.1, 10.1.2.5, 10.2.1.1-5, 10.2.3.1-6, 10.2.4.1-7, 10.2.5.1, 10.2.5.3-7, 10.2.5.9, 10.2.5.11, 10.2.6.1-2, 10.2.7.1-2, 10.2.8.1, 10.2.9.1-3 and 10.2.10.1, the following footnote has been included:

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

On listings 10.1.2.2, 10.1.2.1 and 10.1.2.3, the following column has been included: *Treatment Group\**.

On listings 10.1.2.2, 10.1.2.1 and 10.1.2.3, the following footnote has been included: \*ITZ+LRB/LRB.

On tables 10.2.6.1, 10.2.7.1 and 10.2.8.1 the following footnote has been included: \* Gr 1, Gr 2, Gr 3, Gr 4

#### Section 10.1.1 Patient Disposition

**Original text:** On table 10.1.1.3, the following rows:

Evaluable for PK
Evaluable for Safety

#### Changes to:

#### Included

Evaluable for PK

Evaluable for Safety

#### **Original text:** On table 10.1.1.4, the following header:

| Trot Evaluation for Study 1 art Sequence Subject Reason(s) | Not Evaluable for | Study Part | Sequence | Subject | Reason(s) |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

#### **Changes to:**

| Not Evaluable for | Study Part | Sequence | Subject | Max. Cycle | Reason(s) |
|-------------------|------------|----------|---------|------------|-----------|
| | | | | received | |

### **Original text:** On table 10.1.2.4, the following header:

| Study Part | Sequence | Subject | Reason | Specify |
|------------|----------|---------|--------|---------|

| Study Part | Sequence | Subject | N | Iax, Cycle | received | | Reason | · | | Specify | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Original te | e <u>xt:</u> On tabl | e 10.2.1.1 | , the | follov | ving ro | ows: | | | | | | |
| | | | Par | t A | | Paı | rt B | | Part . | A+B | _ | |
| | | _ | S1 ( | TR) | S1 (T | ΓR) | S2 ( | (RT) | S1 ( | TR) | То | otal |
| | | | N | % | N | % | N | % | N | % | N | 9/ |
| Gender<br>Male<br>Female | | | | | | | | | | | | |
| lace<br>White<br>Black<br>Asian | | | | | | | | | | | | |
| <br>Other (Specify | 7) | | | | | | | | | | | |
| | these two c | lifferent | follo | wing 1 | tables: | | | | | | | |
| | | | Par | t A | | Pai | rt B | | Part | A+B | <b>-</b> т. | .+a1 |
| | | | S1 ( | TR) | S1 (7 | ΓR) | S2 ( | (RT) | S1 ( | TR) | 10 | otal |
| | | | | | | | | % | | | | |

| | Par | t A | | Pai | rt B | | Part | A+B | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | S1 ( | S1 (TR) | | S1 (TR) | | (RT) | S1 (TR) | | Total | |
| | N | % | N | % | N | % | N | % | N | % |
| Race<br>White<br>Black<br>Asian | | | | | | | | | | |
| <br>Other (Specify) | | | | | | | | | , | |

Female

#### (\*\*) Appendix II (Safety Analysis)

#### All Sections

On tables 11.1.1.1-3, 11.1.2.1-2, 11.1.3.1, 11.2.1.1, 11.2.1.2-5, 11.2.1.8, 11.2.1.9, 11.3.1.1-8, 11.3.2.1, 11.4.1.1, 11.4.1.4, 11.4.2.1, 11.4.2.4, 11.4.3.1-4 and 11.7.1.1-3, the following footnote has been included:

Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

On tables and listings 11.1.2.3, 11.1.3.2, 11.1.4.1-3, 11.2.1.10-12, 11.3.1.9, 11.3.2.2, 11.4.1.2-3, 11.4.1.5-6, 11.4.2.2-3, 11.4.2.5-6, and 11.6.2.6 the following column has been included:

#### Treatment Group\*.

On tables and listings 11.1.2.3, 11.1.3.2, 11.1.4.1-3, 11.2.1.10-12, 11.3.1.9, 11.3.2.2, 11.4.1.2-3, 11.4.1.5-6, 11.4.2.2-3, 11.4.2.5-6, and 11.6.2.6 the following footnote has been included:

#### \* ITZ+LRB / LRB.

On tables and listings 11.2.1.2-4, 11.2.1.8, 11.3.1.1-3, 11.3.1.7, 11.4.1.1-3, 11.4.2.1-3 the title:

Worst grade per patient.

Changes to:

Worst grade by treatment.

On tables and listings 11.2.1.5-7, 11.2.1.9, 11.3.1.4-6, 11.3.1.8, 11.4.1.4-6, 11.4.2.4-6 the title:

Worst grade per cycle.

Changes to:

Worst grade per patient.

#### Section 11.2.1 Display of Adverse Events

#### **Original text:** On table 11.2.1.1, the following header:

| | Par | t A | | Pa | rt B | | Part | A+B | | |
|---|---|---|---|---|---|---|---|---|---|---|
| · | S1 ( | TR) | S1 ( | (TR) | S2 - | (RT) | S1 <del>(</del> | TR) | To | otal |
| - | N | % | N | % | N | % | N | % | N | % |

#### **Changes to:**

| Par | t A | | Part B | | |
|------|------|------|--------|------|------|
| S | S1 | | S1 | | 2 |
| Т | R | T | R | R | T |
| N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| Part | A+B | |
|------|------|-------|
| S | 51 | Total |
| T | R | |
| N(%) | N(%) | N(%) |

#### **Original text:** On table 11.2.1.1, the duplicated rows:

No. of patients with dose interruptions associated with treatment-related  $^{\dagger}\ AEs$ 

No. of patients with dose interruptions associated with treatment-related  $\dagger$  AEs

#### **Changes to:**

No. of patients with dose interruptions associated with treatment-related  $^{\dagger}\ AEs$ 

#### The following text has been added: Below table 11.2.1.1:

Supplementary tables describing the adverse event toxicity grades or laboratory abnormality grades 1,2,3,4,5 and grade 1-5 will be added below the tables with aggregated severity grades show in sections 11.2.1, 11.3.1, 11.4.1 and 11.4.2 as shown in table 11.2.1.2

## **Original text:** On table 11.2.1.2 the following header:

| | | P | art A | | | Part B | | | Part A+l | B |
|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | | | | | | | | | Total |
| | | S1 | (TR) | 5 | S1 <del>(TR)</del> | | S2 <del>(RT)</del> | | S1 (TR) | ) |
| | All | Gr > 2 | Gr > 1 | All | Gr > 2 | Gr > 1 | All | Cr > 2 | Gr > 1 | All $Gr \ge 3$ $Gr \ge 4$ |
| | grades | Gi ≥ 3 | Ul ≥ 4 | grades | UI ≥ 3 | Ul ≥ 4 | grades | Ol ≥ 3 | Ul ≥ 4 | grades G1 $\geq$ 3 4 |
| | N % | N % | N % | N % | N % | N % | N % | N % | N % | N % N % N % |

| | | | Pa | rt A | | |
|---|---|---|---|---|---|---|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | Gr ≥ 4 |
| 50011 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | | | | Par | t B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | S | 1 | | | | | S | 2 | | |
| | | T | | | R | | | R | | | T | |
| SOC/PT | All grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr ≥ 4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | Part A- | -B ( <b>S1</b> ) | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|
| | | T | | | R | | | | |
| SOC/PT | All grades | Gr≥3 | Gr≥4 | All<br>grades | Gr≥3 | Gr ≥ 4 | All grades | Gr≥3 | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | | | | ъ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Part | t A | | | | | |
| | | | 7 | Γ | | | | | I | 2 | | |
| SOC/PT | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1-<br>5 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| ••• | | | | | | | | | | | | |
| | | | | | | Part B | (S1) | | | | | |
| | | | 7 | Γ | | | I | ₹ | | | | |
| SOC/PT | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1-<br>5 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| ••• | | | | | | | | | | | | |

| | | | | | | Part B | (S2) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | I | ₹ | | | | | 7 | Γ | | |
| SOC/PT | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gı |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N( |
| ••• | | | _ | | | Part A+B (S1) R Gr 1- 5 Gr1 Gr2 Gr3 Gr4 Gr5 | | | | | | |
| | 1 | · / | | | | | | | | | | |
| SOC/PT | Gr1 | Gr2 | Gr3 | Gr4 | Gr5 | Gr 1- 5 | Gr1 | Gr2 | Gr5 | Gı | | |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N( |
| ••• | | | | | | | | | | | | |
| | | | | | | Tot | al | | | | | |
| | G | r1 | G | r2 | G | r3 | Gı | r4 | G | r5 | Gr | 1- 5 |
| SOC/PT | | | | | | | | | | | | |

Notes: Percentage is based on number of patients by study part and sequence, when applicable.

**Original text:** On tables 11.2.1.3-5, 11.2.1.8, 11.3.1.1-3, 11.3.1.7, 11.4.1.1, 11.4.2.1 the following header:

| | : | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | _ | P | art A | | | Part B | | | Part A+B | |
| SOC / PT | | | | | | | | | | Total |
| | | S1 | (TR) | 1 | S1 <del>(TR)</del> S2 <del>(RT)</del> | | | | S1 <del>(TR)</del> | |
| | All | Gr > 3 | Gr > A | All | All $Gr \ge 3$ $Gr \ge 4$ Algrad | | | Gr > 3 | Gr > A | All $Gr > 3$ $Gr \ge$ |
| | grades | UI ≥ 3 | Ol ≥ 4 | grades | OI ≥ 3 | OI ≥ 4 | grades | GI ≥ 3 | $G_1 \ge 4$ | rades G1 ≥ 3 4 |
| | N % | N % | N % | N % | N % | N % | N % | N % | N % N | N % N % N % |

| | | Part A T R | | | | |
|---|---|---|---|---|---|---|
| | | T | | R | | |
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| 500/11 | N(%) | N(%) | N(%) | | | |

| | | P | art B | |
|---|---|---|---|---|
| | S | 1 | | S2 |
| | T | R | R | T |
| SOC/PT | All $Gr \ge 3$ $Gr \ge 4$ | All $Gr \ge 3$ $Gr \ge 4$ | $4 \frac{\text{All grades}}{\text{grades}} \text{ Gr} \ge 3 \text{ Gr} \ge 6$ | $4 \frac{\text{All}}{\text{grades}} \text{ Gr} \ge 3 \text{ Gr} \ge 4$ |

<sup>†</sup> Related to both or lurbinectedin or itraconazole or with unknown relationship. Part A, patients assigned to Sequence 1; Part B, sequence assigned randomly.

S1, Sequence 1; S2, Sequence 2.

T, Test (ITZ+LRB); R, Reference (LRB alone).

#### $N(\%) \quad N(\%) \quad N(\%)$

| | | | Part A- | +B (S1) | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | Т | | | R | | | Total | |
| SOC/PT | All<br>grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | Gr ≥ 3 | Gr≥4 | All grades | $Gr \ge 3$ | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

## Section 11.2.2 Evolution of Signs and Symptoms during the Treatment

## **Original text:** On table 11.2.2.1 the following header:

| | | | | Wors | t grade | per pat | ient dur | ing trea | tment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA PT | Baseline grade | Gra | de 1 | Gra | de 2 | Gra | de 3 | Gra | de 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | | Pai | rt A | | | | |
| | 1 | | | | | | | | | | |
| | 2 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| ••• | 1 | | | | | | | | | | |
| | ••• | | | | | | G4 (TTD | | | | |
| | | | | | | Part B - | S1 (TR | ) | | | |
| ••• | 1 | | | | | | | | | | |
| ••• | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| ••• | 1 | | | | | | | | | | |
| ••• | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |

| | | | | Wors | t grade | per pat | ient dur | ing trea | tment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA PT | Baseline grade | Gra | de 1 | Gra | de 2 | Gra | de 3 | Gra | de 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | I | Part A - | S1 (TR | 3) | | | |
| | 1 | | | | | | | | | | |
| | 2 | | | | | | | | | | |
| | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | | | | | F | Part B - | S1 (TR | R) | | | |
| | 1 | | | | | | | | | | |
| ••• | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | | | | | F | Part B - | S2 (RT | <u>.</u> | | | |
| ••• | 1 | | | | | | | | | | |
| | 1 | | | | | | | | | | |
| | ••• | | | | | | | | | | |

# Section 11.3.1 Serious Adverse Events

# **Original text:** On tables 11.3.1.1-3 and 11.3.1.7 the following header:

| | | | Pa | rt A | | | | | | Par | t B | | | | | Par | t A+ | -В | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC / PT | | | S1 ( | (TR) | | | S | S1 (7 | TR) | | | S2 ( | RT) | | | S1 | (TR | 2) | | ] | Γota | ıl | |
| | All<br>grades | Gr≥ | ≥ 3 | Gr 4 | 1 | A<br>gra | ll<br>des | Gr | ≥ 3 | G | r 4 | | ll<br>des | Gr | ≥ 3 | G | r 4 | A<br>gra | ll<br>des | Gr | ≥ 3 | Gr | 4 |
| | N % | N | % | N S | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | Ν | <u>~</u> |
| | | | | | | | | | | | | | | | | | | | | | | | _ |

| | | | Pa | ırt A | | |
|--------|------------|------------|--------|------------|------------|--------|
| | | T | | | R | |
| SOC/PT | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr ≥ 4 |
| 500/11 | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | | | | | | | Par | t B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 50.11 | | | | S | 1 | | | | | S | 2 | | |
| 50.11 | | | T | | | R | | | R | | | T | |
| N(%) | SOC/PT | All<br>grades | Gr≥3 | Gr≥4 | All grades | Gr≥3 | Gr ≥ 4 | All grades | Gr≥3 | Gr ≥ 4 | All grades | Gr≥3 | Gr≥4 |
| | | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

| | | | Part A- | +B ( <b>S1</b> ) | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | Т | | | R | | | Total | |
| SOC/PT | All<br>grades | Gr ≥ 3 | Gr ≥ 4 | All grades | Gr≥3 | Gr ≥ 4 | All grades | $Gr \ge 3$ | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |
| | | <u> </u> | <u> </u> | | · · | | | | |

# Section 11.4.1 Hematological Abnormalities

## **Original text:** On tables 11.4.1.1 the following content:

| | | | | P | art 1 | ١ | | | | | Par | t B | | | | | Par | t A+ | -В | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | | | | | | | _ | Tot | al |
| | | | | S1 | (TI | ₹) | | S | S1 (T | TR) | | | S2 ( | RT) | | | S1 | (TR | 2) | | | |
| | Al<br>grad | | Gr | ≥ 3 Gr 4 gr | | A<br>gra | ll<br>des | Gr | ≥ 3 | G | r 4 | | ll<br>des | Gr | ≥ 3 | G | r 4 | All<br>grad | | 6r ≥ 3 | 3 Gr 4 | |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N ' | % ] | N % | N % |
| Anemia | | | | | | | | | | | | | | | | | | | | | | |
| Leukopenia | | | | | | | | | | | | | | | | | | | | | | |
| Lymphopenia | | | | | | | | | | | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | | | | | | | | | | | |
| Thrombocytopenia | | | | | | | | | | | | | | | | | | | | | | |

## **Changes to:**

| | | | | | | Par | t A | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <del></del> | | 7 | Γ | | | | | F | ₹ | | |
| SOC/PT | All gra | des | Gr | ≥ 3 | Gr | ≥4 | All g | rades | Gr | ≥ 3 | Gr | ≥4 |
| 50011 | N(%) | ) | N( | %) | N( | %) | N( | %) | N( | %) | N( | %) |
| Anemia<br>Leukopenia<br>Lymphopenia<br>Neutropenia<br>Fhrombocytopenia | | | | | | | | | | | | |
| | | | | | | Pai | rt B | | | | | |
| | | | S | 1 | | | | | S | 2 | | |
| | | T | | | R | | | R | | | T | |
| SOC/PT | All<br>grades G | ir≥3 | Gr ≥ 4 | All<br>grades | $Gr \ge 3$ | Gr ≥ 4 | All<br>grades | $Gr \ge 3$ | Gr ≥ 4 | All<br>grades | $Gr \ge 3$ | Gr≥ |
| | N(%) N | V(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(% |
| Anemia<br>Leukopenia<br>Lymphopenia<br>Neutropenia<br>Thrombocytopenia | | | | | | | | | | | | |
| | | | Part A+ | B (S1) | | | | | T | otal | | |
| | Т | , | | | R | | | | | | | |

| | | | Part A- | +B (S1) | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | Т | | | R | | | Total | |
| SOC/PT | All grades | Gr≥3 | Gr ≥ 4 | All grades | Gr≥3 | Gr≥4 | All grades | $Gr \ge 3$ | Gr≥4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

Anemia Leukopenia Lymphopenia Neutropenia Thrombocytopenia

## Section 11.4.2 Biochemical Abnormalities

# **Original text:** On tables 11.4.2.1 the following content:

| | | | P | art A | 4 | | | | | Par | tΒ | | | | | Par | t A+ | В | _ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | S | l (TI | R) | | 9 | S1 (T | R) | | | S2 ( | RT) | | | S1 | (TR | .) | | То | tal |
| | All<br>grade | Gr | ≥ 3 | G | r 4 | A<br>gra | dl<br>des | Gr | ≥3 | Gı | r 4 | | ll<br>des | Gr | ≥ 3 | G | r 4 | A<br>grad | | Gr≥ | 3 Gr 4 |
| | N % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N % | 6 N % |
| ALT increase<br>AST increase<br>* | | | | | | | | | | | | | | | | | | | | | |

## **Changes to:**

| | | | | | | Par | t A | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | , | Т | | | | R | |
| | A | ll grades | Gr | ≥ 3 | Gr | ≥ 4 | All grades | Gr≥3 | Gr ≥ 4 |
| | | N(%) | N( | (%) | N( | %) | N(%) | N(%) | N(%) |
| ALT increase<br>AST increase<br>* | | | | | | | | | |
| | | | | | | Par | t B | | |
| | | | S | S1 | | | | S2 | |
| | | Т | | | R | | R | | T |
| | Al<br>grad | | 3 Gr≥4 | All<br>grades | $Gr \ge 3$ | Gr ≥ 4 | $\frac{\text{All grades}}{\text{grades}} \text{ Gr} \ge 3$ | 3 Gr≥4 All<br>grade | $Gr \ge 3 Gr \ge$ |
| | N(% | %) N(% | ) N(%) | N(%) | N(%) | N(%) | N(%) N(%) | N(%) N(%) | ) N(%) N(% |
| ALT increase<br>AST increase<br>* | | | , | | | | | | |
| | :: | | Part A+ | -R (\$1) | | | | | |
| | | T | T uit 71 | <i>B</i> (51) | R | | _ | Total | |
| | All<br>grades | $Gr \ge 3$ | Gr≥4 | All grades | Gr≥3 | Gr≥4 | 4 All grades | $Gr \ge 3$ | Gr ≥ 4 |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) |

AST increase

# Section 11.4.3 Laboratory Values Over Treatment

**Original text:** On table 11.4.3.1 the following content:

| | | | | Wors | t grade | per pat | ient dur | ing trea | tment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline grade | Gra | de 1 | Gra | de 2 | Gra | de 3 | Gra | de 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | | Pa | rt A | | | | |
| Anemia | 0 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| Leukopenia | 0 | | | | | | | | | | |
| | <br>4 | | | | | | | | | | |
| | 0 | | | | | | | | | | |
| ••• | | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| | | | | | ] | Part B - | S1 (TR | (1) | | | |
| Anemia | 0 | | | | | | | | | | |
| memia | | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| Leukopenia | 0 | | | | | | | | | | |
| | 4<br>0 | | | | | | | | | | |
| ••• | | | | | | | | | | | |
| | <br>4 | | | | | | | | | | |
| | <u>'</u> | | | | | | | | | | |
| Anemia | 0 | | | | | • | •• | | | | |
| Michila | | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| Leukopenia | 0 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| ••• | 0 | | | | | | | | | | |
| | 4 | | | | | | | | | | |

| | | | | Wors | st grade | per pa | tient dur | ing trea | atment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline grade | Gra | de 1 | | de 2 | | ade 3 | | ide 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | ] | Part A | - S1 (TR | 3) | | | |
| Anemia | <b>G</b> 0 | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| Leukopenia | $\mathbf{G}0$ | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| ••• | $\mathbf{G}0$ | | | | | | | | | | |
| | <b>G</b> 4 | | | | | 5 . 5 | G4 (TTP) | | | | |
| | н | | | | - | Part B | - S1 (TR | .) | | | |
| Anemia | $\mathbf{G}0$ | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | G4 | | | | | | | | | | |
| Leukopenia | $\mathbf{G}0$ | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | G4 | | | | | | | | | | |
| ••• | $\mathbf{G}0$ | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| | | | | | ] | Part B | - S2 (RT | <u>()</u> | | | |
| Anemia | $\mathbf{G}0$ | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| Leukopenia | $\mathbf{G}0$ | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| ••• | $\mathbf{G}0$ | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |

# **Original text:** On table 11.4.3.3 the following content:

| | | | | Wors | st grade | per pat | ient dur | ing trea | tment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline grade | Gra | de 1 | | de 2 | | de 3 | | de 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | | Pa | rt A | | | | |
| ALT increase | 0 | | | | | | | | | | |
| | <br>4 | | | | | | | | | | |
| AST increase | 0 | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| | 0 | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| | | | | | ] | Part B - | S1 (TR | .) | | | |
| ALT increase | 0 | | | | | | | <i>)</i> | | | |
| A COTT : | 4 | | | | | | | | | | |
| AST increase | 0 | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| | 0 | | | | | | | | | | |
| | 4 | | | | | | | | | | |
| | | | | | | | •• | | | | |
| ALT increase | 0 | | | | | | | | | | |
| | <br>4 | | | | | | | | | | |
| AST increase | 0 | | | | | | | | | | |
| | 4<br>0 | | | | | | | | | | |
| ••• | | | | | | | | | | | |
| | 4 | | | | | | | | | | |

| | | | | Wors | st grade | per pa | tient dur | ing trea | atment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline grade | Gra | de 1 | | de 2 | | ide 3 | | ide 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | ] | Part A - | - S1 (TR | 3) | | | |
| ALT increase | <b>G</b> 0 | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| AST increase | $\mathbf{G}0$ | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| | $\mathbf{G}0$ | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| | | | | | - | Part B | - S1 (TR | .) | | | |
| ALT increase | $\mathbf{G}0$ | | | | | | | | | | |
| | G4 | | | | | | | | | | |
| AST increase | $\mathbf{G}0$ | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | G4 | | | | | | | | | | |
| | $\mathbf{G}0$ | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| | | | | | I | Part B | - S2 (RT | [) | | | |
| ALT increase | $\mathbf{G}0$ | | | | | | | | | | |
| | G4 | | | | | | | | | | |
| AST increase | $\mathbf{G}0$ | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | <b>G</b> 4 | | | | | | | | | | |
| ••• | $\mathbf{G}0$ | | | | | | | | | | |
| | <b>G</b> 4 | _ | | | | | | | | | |

# Section 11.6.1 Physical Findings, ECOG PS

# **Original text:** On listings 11.6.1.1-3, 11.6.2.2-5 the following content:

| Study p | art / Sequence | Subject |
|---------|----------------|---------|
| Part A | | |
| Part B | S1 (TR) | |
| | S2 (RT) | |

| Study p | art / Sequence | Treatment<br>Group* | Subject |
|---------|----------------|---------------------|---------|
| Part A | S1 (TR) | | ••• |
| Part B | S1 (TR) | | |
| | S2 (RT) | | |

## Section 11.6.2 LVEF and ECG

### **Original text:** On listings 11.6.2.2 the following header:

| Study nort / | | PR interval | | % Chai | nge <sup>†</sup> | |
|---|---|---|---|---|---|---|
| Study part / Sequence | Subject | (msec) <sup>‡</sup> at baseline | Cycle 1<br>Pre infusion | Cycle 1<br>Post infusion | | ЕОТ |

#### **Changes to:**

| G. 1 / | - | PR interval | | % Change <sup>†</sup> | |
|---|---|---|---|---|---|
| Study part / | Subject | (msec) <sup>‡</sup> at | Cycle 1 | Cycle 2 | EOT |
| Sequence | | baseline | Pre infusion Post infusion | Pre infusion Post infusion | EOT |

### **Original text:** On listings 11.6.2.3 the following header:

| Study part / | | Haart rata (hnm)‡ | | % Ch | iange <sup>†</sup> | |
|---|---|---|---|---|---|---|
| Sequence Sequence | Subject | Heart rate (bpm) <sup>‡</sup> at baseline | Cycle 1 | Cycle 2<br>Pre infusion | Cycle 2<br>Post infusion | ЕОТ |

#### **Changes to:**

| C4- 1 / | | Heart rate | | % Change <sup>†</sup> | |
|---|---|---|---|---|---|
| Study part / | Subject | (bpm) <sup>‡</sup> | Cycle 1 | Cycle 2 | ЕОТ |
| Sequence | _ | at baseline | <b>Pre infusion Post infusion</b> | Pre infusion Post infusion | EUI |

### **Original text:** On listings 11.6.2.4 the following header:

| Study part / | | OT interval (msec) <sup>‡</sup> | | % Cł | iange <sup>†</sup> | |
|---|---|---|---|---|---|---|
| Sequence Sequence | Subject | at baseline | Cycle 1 | Cycle 2<br>Pre infusion | Cycle 2<br>Post infusion | ЕОТ |

### Changes to:

| C4 1 / | | QT interval | | % Change <sup>†</sup> | |
|---|---|---|---|---|---|
| Study part /<br>Sequence | Subject | (msec) <sup>‡</sup> | Cycle 1 | Cycle 2 | ЕОТ |
| Sequence | | at baseline | <b>Pre infusion Post infusion</b> | Pre infusion Post infusion | EOI |

## **Original text:** On listings 11.6.2.5 the following header:

| Study part / | | OTc (Bazett's)‡ | | % Cł | nange <sup>†</sup> | |
|---|---|---|---|---|---|---|
| Sequence Sequence | Subject | at baseline | Cycle 1 | Cycle 2<br>Pre infusion | Cycle 2<br>Post infusion | ЕОТ |

| Study part / QTc (Bazett's) <sup>‡</sup> Cycle 1 Cycle 2 | |
|----------------------------------------------------------|-----|
| Sequence at baseline Cycle 2 | EOT |
| Pre infusion Post infusion Pre infusion Post infusion | EOI |

# **Original text:** On listings 11.6.2.6 the following header:

| Study Sequence | Subject Assessment | Visit | ECG# | Result Specify | PR | Heart | QT | QTc <sup>†</sup> |
|---|---|---|---|---|---|---|---|---|
| Part | date | | | | interval | rate | interval | (Bazett's) |
| | | | | | (msec) | (bpm) | (msec) | |

| StudySequence 7 | Treatment Subject | Cycle Assess | m Visit | ECG #‡ | Result | Specify | PR | Heart | QT | QTc <sup>†</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Part | Group* | ent da | te | | | | interval | rate | interval | (Bazett' |
| | | | | | | | (msec) | (bpm) | (msec) | s) |

## Section 11.7.1 Concomitant medication during treatment (ATC1/ATC2/ATC4/PN)

### **Original text:** On table 11.7.1.1 the following header:

| Paı | t A | | Pa | rt B | | Part | A+B | | |
|---|---|---|---|---|---|---|---|---|---|
| S1 (TR) | | S1 ( | (TR) | S2 | S2 (RT) | | S1 (TR) | | Total |
| 51 ( | 110) | 51 ( | (TR) | 52 | (1(1) | 51 ( | 11() | | _ |
| <br>N | % | N | % | N | % | N | % | N | % |

## **Changes to:**

| Part A | | | Part B | | | Part A+B(S1) | | |
|---|---|---|---|---|---|---|---|---|
| T | R | T | R | Т | R | T | R | |
| N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |

# **Original text:** On listings 11.7.1.2 the following header:

| Part A | | Part A Part B | | | | | A+B | _ | |
|--------|-----|---------------|------|------|------|------|-----|----|------|
| S1 ( | TR) | S1 ( | (TR) | S2 ( | (RT) | S1 ( | TR) | To | otal |
| N | % | N | % | N | % | N | % | N | % |

| Pai | t A | | Part B | | | | Part A+B (S1) | |
|---|---|---|---|---|---|---|---|---|
| Т | R | T | R | T | R | T | R | Total |
| N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |

# **Original text:** On listings 11.7.1.3 the following header:

| Part A | Pai | rt B | Part A+B | _ |
|---------|---------|---------|----------|-------|
| | | | | Total |
| S1 (TR) | S1 (TR) | S2 (RT) | S1 (TR) | |

| Par | t A | A Part B Part A+B (S1) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| T | R | T | R | T | R | T | R | Total |
| N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |

## (\*\*\*) Appendix IV (DB Listings)

#### All Sections

On listings 13.6, 13.7, 13.12, 13.16, 13.17, 13.19-36, 13.42 from Appendix IV the following footnote has been included:

\* ITZ+LRB / LRB.

Also on the same listings from Appendix IV the following column has been included: *Treatment Group\**.

Column Cycle, has been included also on these listings, where applicable.